

### CLINICAL STUDY PROTOCOL

Study Title: A Phase 2, Open-Label, Multicenter, Multi-cohort, Single-Arm

Study to Investigate the Safety and Efficacy of Sofosbuvir + Ribavirin in Adolescents and Children with Genotype 2 or 3

Chronic HCV Infection

Sponsor: Gilead Sciences, Inc.

333 Lakeside Drive

Foster City, CA 94404, USA

IND No.: 106,739 EudraCT Number: TBD

Indication: Hepatitis C Virus Infection

Protocol ID: GS-US-334-1112

Gilead Sciences Medical

: Telephone:

Monitor:

Name: Luisa Stamm, MD, PhD
Telephone: PPD

Mobile: PPD

Fax: PPD

E-mail: PPU

Protocol Version/Date: Original: 20 December 2013

### CONFIDENTIALITY STATEMENT

The information contained in this document, particularly unpublished data, is the property or under control of Gilead Sciences, Inc., and is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Institutional Review Board or Independent Ethics Committee. The information is only to be used by you in connection with authorized clinical studies of the investigational drug described in the protocol. You will not disclose any of the information to others without written authorization from Gilead Sciences, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

# TABLE OF CONTENTS

| TA | BLE O | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF I | N-TEXT FIGURES | 4 |
| PRO | OTOCO | OL SYNOPSIS | 5 |
| GL | OSSAR | RY OF ABBREVIATIONS AND DEFINITION OF TERMS | 14 |
| 1. | INTRODUCTION | | |
| | 1.1. | Background | 17 |
| | 1.2. | Sofosbuvir | |
| | 1.3. | Ribavirin (RBV) | |
| | 1.4. | Rationale for the Current Study | |
| | 1.5. | Rationale for Dose Selection of SOF | |
| | 1.6. | Overall Risk/Benefit Assessment | 20 |
| 2. | OBJE | ECTIVES | 22 |
| 3. | STUI | DY DESIGN | 23 |
| | 3.1. | Treatment Plan and Regimen | |
| | | 3.1.1. Part A | |
| | | 3.1.2. Part B | |
| | 3.2. | Visit Schedule | |
| | | 3.2.1. Part A | |
| | 2.2 | 3.2.2. Part B | |
| | 3.3.<br>3.4. | Virologic Response-Based Stopping Criteria. | |
| | 3.4. Treatment Discontinuations Criteria 3.5. Discontinuations | | |
| | 3.6. | Pharmacogenomic Substudy | |
| | 3.7. Long Term Follow Up | | |
| 4. | SUBJECT POPULATION | | |
| | 4.1. | Number of Subjects and Subject Selection | 28 |
| | 4.2. | Inclusion Criteria | 28 |
| | 4.3. | Exclusion Criteria | 28 |
| 5. | INVESTIGATIONAL MEDICINAL PRODUCTS3 | | |
| | 5.1. Randomization and Blinding. | | |
| | 5.2. | Sofosbuvir | |
| | | 5.2.1. Description and Handling | 30 |
| | | 5.2.2. Storage and Handling | |
| | | 5.2.3. Dosage and Administration of SOF | |
| | 5.3. | Ribavirin | |
| | | 5.3.1. Description and Handling of RBV | |
| | E 1 | 5.3.2. Dosage and Administration of RBV | |
| | 5.4.<br>5.5. | | |
| | | 5.6. Prior and Concomitant Medications. | |
| 6. | STUDY PROCEDURES | | |
| 0. | | | |
| | 6.1.<br>6.2. | Subject Enrollment | |
| | 0.2. | 6.2.1. Screening Visit (Day –28 to Day 0) | |
| | | 5.2.1. Solotining visit (Day 20 to Day 0) | |

| | 6.3. | Part A: 7 | Treatment Assessments | 37 |
|---|---|---|---|---|
| | | 6.3.1. | Day 1 Visit | |
| | | 6.3.2. | Day 3 | 38 |
| | | 6.3.3. | Day 7 – Intensive PK | 38 |
| | 6.4. | Part B: 7 | Treatment Assessments | 40 |
| | | 6.4.1. | Day 1 Visit | 40 |
| | | 6.4.2. | Weeks 1 and 2 (± 3 days) | 41 |
| | | 6.4.3. | Weeks 4 and 8 (± 3 days) | 42 |
| | | 6.4.4. | Week 12 (± 3 days) | |
| | | 6.4.5. | Week 16 and 20 (± 3 days) – GT-3 Subjects only | |
| | | 6.4.6. | Week 24(± 3 days) – GT-3 Subjects only | |
| | | 6.4.7. | Unscheduled Visit/Early Termination Visit | |
| | 6.5. | Post-Tre | atment Assessments | |
| | | 6.5.1. | 4-Week Post-Treatment Visit (± 5 days) | |
| | | 6.5.2. | 12-Week Post-Treatment Visit (± 5 days) | |
| | | 6.5.3. | 24-Week Post-Treatment Visit (± 5 days) | |
| | 6.6. | | res and Specifications. | |
| | 0.0. | 6.6.1. | Clinical Laboratory Analytes | |
| | | 6.6.2. | Medical History | |
| | | 6.6.3. | Complete Physical Examination | |
| | | 6.6.4. | Tanner Pubertal Stage Assessment. | |
| | | 6.6.5. | Vital Signs | |
| | | 6.6.6. | Body Mass Index (BMI) | |
| | | 6.6.7. | Viral Sequencing (Archive) | |
| | | 6.6.8. | | |
| | | 6.6.9. | Pregnancy Testing | 49 |
| 7. | TOXI | CITY MA | NAGEMENT | |
| | 7.1. | Modifies | ation of Dose/Schedule Due to Toxicity | 50 |
| | 7.1. | 7.1.1. | RBV Dose Adjustments | |
| | 7.2. | | Stopping Rules for SOF | |
| _ | | _ | | |
| 8. | ADVERSE EVENTS MANAGEMENT | | | |
| | 8.1. | Definition | ons of Adverse Events, Adverse Reactions, and Serious Adverse Events | 51 |
| | | 8.1.1. | Adverse Events. | |
| | | 8.1.2. | Serious Adverse Events | 51 |
| | | 8.1.3. | Clinical Laboratory Abnormalities and Other Abnormal Assessments | |
| | | | as Adverse Events or Serious Adverse Events | 52 |
| | 8.2. | Assessm | ent of Adverse Events and Serious Adverse Events | |
| | | 8.2.1. | Assessment of Causality for Study Drugs and Procedures | |
| | | 8.2.2. | Assessment of Severity | 53 |
| | 8.3. | | ator Requirements and Instructions for Reporting Adverse Events and Serious | |
| | | | Events | |
| | 8.4. | | Reporting Requirements | |
| | 8.5. | | Situations Reports | |
| | | 8.5.1. | Definitions of Special Situations | |
| | | 8.5.2. | Instructions for Reporting Special Situations | 56 |
| 9. | STAT | TISTICAL | CONSIDERATIONS | 58 |
| | 9.1. | Analysis | Objectives and Endpoints | |
| | | 9.1.1. | Analysis Objectives | |
| | | 9.1.2. | Primary Endpoint | |
| | | 913 | Secondary Endpoints | 50 |

| | Figure | 3-1. | Study Schema | 25 |
|---|---|---|---|---|
| | | | LIST OF IN-TEXT FIGURES | |
| | | | rotential, and Contraceptive Requirements | 105 |
| | Apper | iaix 5. | Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements | 105 |
| | Appendix 4. Appendix 5. | | Tanner Stages | 104 |
| | | | Laboratory Abnormalities | |
| | Appendix 3. | | GSI Grading Scale for Severity of Adverse Events and | |
| | Apper | dix 2. | Study Procedures Table | |
| | Apper | | Investigator Signature Page | |
| 12. | | | | |
| 11. | REFE | RENCES . | | 72 |
| | | 10.3.3. | Study Discontinuation | |
| | | 10.3.2. | Access to Information for Auditing or Inspections | |
| | | 10.3.1. | Access to Information for Monitoring. | |
| | 10.3. | | vestigator/Sponsor Responsibilities | |
| | 10.2 | 10.2.2. | Study Report and Publications | |
| | | 10.2.1. | Protocol Modifications | |
| | 10.2. | - | Responsibilities | |
| | 10.5 | 10.1.9. | Protocol Compliance | |
| | | 10.1.8. | Inspections | |
| | | 10.1.7. | Drug Accountability | |
| | | 10.1.6. | Case Report Forms | |
| | | 10.1.5. | Study Files and Retention of Records | |
| | | 10.1.4. | Confidentiality | |
| | | 10.1.3. | Informed Consent/Assent | 67 |
| | | | (IEC) Approval. | |
| | | 10.1.2. | Institutional Review Board (IRB)/Independent Ethics Committee | |
| | | 10.1.1. | | |
| | 10.1. | Investiga | ator Responsibilities | 66 |
| 10. | RESP | ONSIBILI | TIES | 66 |
| | | • | | |
| | 9.7.<br>9.8. | | Size | |
| | 9.7. | | onitoring Committee | |
| | | 9.6.3.<br>9.6.4. | Other Safety Evaluations | |
| | | 9.6.2.<br>9.6.3. | Laboratory Evaluations | |
| | | 9.6.1.<br>9.6.2. | Extent of Exposure | |
| | 9.6. | 9.6.1. | Inalysis | |
| | 0.6 | 9.5.3. | Subgroup Analysis | |
| | | 9.5.2. | Secondary Analysis | |
| | | 9.5.1. | Primary Analysis | |
| | 9.5. | | Analysis | |
| | 9.4. | | cokinetic Analysis | |
| | 9.3. | | aphic Data and Baseline Characteristics | |
| | | 9.2.3. | Interim Analysis | |
| | | 9.2.2. | Data Handling Conventions | |
| | | 9.2.1. | Analysis Sets | |
| | 9.2. | Analysis | s Conventions | 59 |

# PROTOCOL SYNOPSIS Gilead Sciences, Inc. 333 Lakeside Drive Foster City, CA 94404, USA

| Study Title: | A Phase 2, Open-Label, Multicenter, Multi-cohort, Single-Arm<br>Study to Investigate the Safety and Efficacy of Sofosbuvir +<br>Ribavirin in Adolescents and Children with Genotype 2 or 3<br>Chronic HCV Infection |
|---|---|
| IND Number: | 106,739 |
| <b>EudraCT Number:</b> | TBD |
| Study Centers: | Approximately 50 sites in the United States, Europe, Russia, Australia, and New Zealand |
| Number of Subjects: | Approximately 100 subjects |
| Target Population: | Adolescents and children (aged 3 to < 18) with chronic hepatitis C virus (HCV) infection |
| <b>Treatment Duration:</b> | Part A – 7 days |
| | Part B – 12 or 24 weeks |

# **Objectives:**

The primary objective of Part A of this study is:

 To evaluate the steady state pharmacokinetics (PK) and confirm the dose of sofosbuvir (SOF) in HCV-infected pediatric subjects

The secondary objective of Part A of this study is:

 To evaluate the safety and tolerability of 7 days of dosing of SOF in HCV-infected pediatric subjects

The primary objectives of Part B of this study are:

- To evaluate the safety and tolerability of SOF + ribavirin (RBV) for 12 or 24 weeks in HCV-infected pediatric subjects with genotype 2 or 3, respectively
- To determine the antiviral efficacy of SOF+RBV treatment in genotype 2 and genotype 3 HCV-infected subjects separately, as assessed by the proportion of subjects with SVR 12 weeks after completion of treatment (SVR12)

The secondary objectives of Part B of this study are:

- To determine the antiviral efficacy of SOF+RBV treatment in genotype 2 and genotype 3 HCV-infected subjects separately, as assessed by the proportion of subjects with SVR 4 and 24 weeks after completion of treatment (SVR4 and SVR24)
- To evaluate the kinetics of circulating HCV RNA during treatment and after completion of treatment
- To evaluate the emergence of viral resistance to SOF during treatment and after completion of treatment

The exploratory objective of this study is:

PPD

### Study Design:

Open-label, multi-cohort, two-part study evaluating the PK, safety, and antiviral activity of SOF in chronic HCV-infected pediatric subjects.

The study will be divided into 2 parts as follows:

<u>Part A</u>: Part A (PK lead-in) will evaluate and/or confirm age appropriate SOF doses by analyzing PK, safety, and antiviral activity of SOF through 7 days of dosing for each of three cohorts. Children aged 3 to 6, children aged 6 to < 12 years and adolescents aged 12 to < 18 years with genotype (GT) 2 or 3 HCV infection and evidence of HCV RNA > 1000 IU/mL at study entry will be evaluated.

Three cohorts of up to 10 subjects each will be sequentially enrolled:

- Cohort 1: 12 to < 18 years old weighing  $\ge$  45kg
- Cohort 2: 6 to < 12 years old</li>
- <u>Cohort 3:</u> 3 to < 6 years old</li>

The study will start with Cohort 1. Subjects will receive SOF (400-mg adult tablet or 4 x 100-mg tablets if determined necessary based on SOF swallowability assessment) for 7 days with intensive PK conducted on Day 7.

Subjects in each cohort (Cohorts 1, 2 and 3) will immediately enroll in Part B as they complete Day 7 of Part A. They will begin dosing with SOF + RBV with no interruption of study drug administration.

Following completion of study treatment in Cohort 1 (Part A) and pending PK and safety results from Cohort 1 (Part A), Cohort 2 will initiate and receive study treatment (age-appropriate formulation). Following completion of study treatment in Cohort 2 (Part A) and pending PK and safety results from Cohort 2 (Part A), Cohort 3 will receive study treatment (age-appropriate formulation).

**Part B**: Part B will be initiated by dose cohort after confirmation of age-appropriate SOF dosage levels. Subjects who participated in Part A will immediately rollover into Part B (Day 1), with no interruption of study drug administration:

Children aged 3 to < 12 years and adolescents aged 12 to < 18 years with GT-2 or GT-3 infection and evidence of HCV RNA > 1000 IU/mL at study entry (those who were dosed in Part A will have met this criteria prior to enrollment) will be evaluated.

Subjects enrolled in Part B will receive the following regimen.

- GT-2 subjects: SOF + RBV for 12 weeks
- GT-3 subjects: SOF + RBV for 24 weeks

The study will enroll both treatment-naïve and treatment-experienced pediatric subjects, with up to 20 subjects allowed to be treatment experienced. Approximately 100 total subjects, including subjects from Part A, will be enrolled in Part B as follows

- Group 1: Approximately 50 adolescent subjects (12 to < 18 years of age)
- Group 2: Approximately 50 pediatric subjects (3 to < 12 years of age)

The following definitions will be used for treatment-experienced subjects:

- <u>Interferon intolerant:</u> Subject who discontinued therapy (≤ 12 weeks total) due to ≥ 1 adverse event
- <u>Interferon non-responder:</u> Subject who did not achieve undetectable HCV RNA levels while on treatment
- <u>Relapse/breakthrough:</u> Subject who achieved undetectable HCV RNA during treatment or within 4 weeks of the end of treatment but did not achieve a sustained virologic response (SVR)

The study schedule contains the following visits: Screening, Day 1, Weeks 1, 2, 4, 8, 12 (and Weeks 16, 20, and 24 for GT-3) during the treatment phase followed by post-treatment visits 4, 12 and 24 weeks after discontinuation of therapy.

All subjects who do not attain SVR or have viral relapse will be encouraged to discuss treatment with standard-of-care (SOC) therapy with their healthcare provider.

Substudy and Long-Term Follow-Up Study:

# Pharmacogenomics (PG) Substudy

PPD

# Long-Term Follow-up

Subjects who attain SVR24 or those who do not attain SVR24 and do not initiate experimental or approved anti-HCV therapy will be followed every 6 months for assessments of growth, quality of life, and long-term viral suppression (if applicable) in a separate protocol. This follow-up will continue for 5 years.

Diagnosis and Main Eligibility Criteria:

Chronic HCV-infected, treatment-naïve and up to 20 subjects may be treatment experienced, male and female subjects aged 3 to < 18.

### Inclusion Criteria:

- Documented chronic GT 2 or 3 HCV infection
- HCV RNA ≥ 1000 IU/mL at Screening
- Part A only: subjects in cohort 1 (age 12 to <18 years of age) must weigh ≥ 45kg
- Agree to use 2 forms of highly effective contraception, as referenced in Appendix 5, for the duration of the study and for 6 months (for female subjects) or 7 months (for male subjects) after the last dose of study medication if age, cultural, and sexual activity status appropriate (eg: if sexually active; does not pertain to pre-pubertal subjects). Females of childbearing potential (as defined in Appendix 5) must have a negative pregnancy test at Screening and Day 1.

### **Exclusion Criteria:**

- Hematologic or biochemical parameters at screening outside the protocol-specified requirements
- HIV, acute hepatitis A virus (HAV) or chronic HBV infection

- Decompensated liver disease
- Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers)
- Chronic liver disease of a non-HCV etiology (eg, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency)
- Chronic use of systemic immunosuppressive agents or immunomodulatory agents
- Active or recent history ( $\leq 1$  year) of drug or alcohol abuse
- History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.

See Sections 4.2 and 4.3 of the protocol for full eligibility criteria.

Study Procedures/ Frequency:

# Part A:

Screening assessments will be completed within 28 days of the Day 1 visit.

Screening assessments will include: physical examination, vital signs (including height and weight), Tanner Pubertal Stage assessment, concomitant medications, safety laboratory tests, coagulation tests, HCV RNA, serology (HIV, HAV, HCV, HBV), alpha-1 anti-trypsin, serum  $\beta$ -human chorionic gonadotropin hCG (females of childbearing potential only), thyroid stimulating hormone, HbA1c, IL28B genotyping, alpha fetoprotein, urinalysis, and urine drug screen.

Study Visits will occur at Screening, Day 1, Day 3, and Day 7

On-Treatment assessments include adverse events (AEs), concomitant medications, physical examination, vital signs, height, weight, safety laboratory tests, HCV RNA, viral sequencing sampling, urine pregnancy tests (females of child bearing potential only), and urinalysis. Coagulation will be performed at Day 1 only. SOF swallowability assessment will be performed on Day 1 for a subject's ability to swallow the 400 mg SOF tablet (only subjects administered SOF in tablet form).

Subjects (up to 10 subjects) enrolled in Part A will participate in an intensive PK evaluation on Day 7. Following completion of the Day 7 intensive PK visit, subjects will then return for scheduled study visits outlined in Part B and begin dosing with SOF + RBV with no interruption of study drug administration.

# Part B:

Screening assessments will be completed within 28 days of the Day 1 visit. For subjects continuing from Part A, screening for Part B will not be required.

Screening assessments will include physical examination, vital signs, concomitant medications, safety laboratory tests, HCV RNA, serology (HIV, HAV, HCV, HBV), alpha-1 anti-trypsin serum  $\beta$ -human chorionic gonadotropin hCG (females of childbearing potential only), thyroid stimulating hormone, IL28B genotyping, urinalysis, and urine drug screen.

- <u>GT-2 Subjects:</u> Study visits for GT-2 subjects will occur at screening, Day 1, and the end of Weeks 1, 2, 4, 8, and 12.
- GT-3 Subjects: Study visits for GT-3 subjects will occur at screening, Day 1, and the end of Weeks 1, 2, 4, 8, 12, 16, 20, and 24.

All Part B subjects will then return for follow-up visits at 4, 12 and 24 weeks after discontinuation of therapy.

On-treatment assessments will include adverse events, concomitant medications, physical examination, vital signs (including height and weight), safety laboratory tests, coagulation tests, HCV RNA, PK samples, and urine pregnancy tests (females of childbearing potential only). Rates of growth (height and weight percentiles) and Tanner Pubertal Stage assessment will be assessed at Day 1, end of treatment, post-treatment Week 12 and at the end of the 24-week follow-up phase; parental heights will be recorded at Day 1. When available, results from liver biopsies performed within 2 years prior to screening will be collected at Day 1. SOF swallowability assessment will be performed on Day 1 for a subject's ability to swallow the 400 mg SOF tablet (all subjects administered SOF in tablet form).

Post-treatment assessments will include adverse events, concomitant medications, vital signs, safety laboratory tests, HCV RNA, and urine pregnancy tests (females of childbearing potential only). Samples for viral RNA sequencing/phenotyping will be collected at Day 1 and every visit thereafter.

PPD

CONFIDENTIAL Page 10 20 December 2013

# Test Product, Dose, and Mode of Administration:

# Age group 12 to < 18 years:

Part A: (Cohort 1) SOF 400-mg tablets will be administered once daily. Subjects determined unable to swallow the 400-mg tablet (by SOF swallowability assessment at Day 1 or at any time during the study) will be re-assigned to 4 x 100-mg tablets daily. Subjects who weigh <45 kg are excluded from this age group in Part A.

Part B: SOF 400-mg tablets will be administered once daily for subjects who weigh  $\geq$  45 kg. Subjects determined unable to swallow the 400-mg tablet (by SOF assessment at Day 1 or at any time during the study) will be re-assigned to 4 x 100-mg tablets daily. For subjects in this age group who weigh < 45 kg, PK data from part A will be used to determine the appropriate dose of SOF to be administered.

Subjects who participated in Part A will continue the assigned dose in Part B.

# Age group 3 to < 12 years:

(Part A and Part B) SOF age-appropriate formulation will be administered once daily with a dose and formulation to be determined.

# **RBV Weight-Based Dosing (All age groups):**

The RBV dose is:

- 15 mg/kg divided BID for subjects with weight below 50 kg
- 400 mg BID for subjects weighing  $\geq$  50 to less than 65 kg
- 400 mg q AM and 600 mg q PM (i.e., 1,000 mg Total Daily Dose) for subjects weighing ≥ 65 kg to less than 75 kg
- 600 mg BID for subjects with weights greater than 75 kg.

The morning dose of RBV will be taken with an age-appropriate dose of SOF with food. The evening dose of RBV will be taken with food.

**Reference Therapy:** 

None

### **Evaluation Criteria:**

Safety: AEs, laboratory tests, and Tanner Pubertal Stage assessments will

be collected throughout the study.

Efficacy: Efficacy will be evaluated using scheduled assessments of HCV

RNA performed using COBAS® AmpliPrep/COBAS® TaqMan®

HCV Test.

PK:

For subjects in Part A, steady-state PK of SOF and its major metabolites GS-566500 and GS-331007 will be assessed at Day 7. For Cohorts 1 and 2, plasma samples will be collected for PK analyses following dosing of study drugs on Day 7 at the following time points: 0 (predose), 0.5, 1, 2, 3, 4, 8, and 12 hours postdose (with predose also serving as t=24). For Cohort 3, plasma samples for PK analyses will be collected at the following time points: 0 (predose), 2, 4, 8, and 12 hours postdose (with predose also serving as t=24).

Plasma PK parameters such as  $C_{max}$ ,  $T_{max}$ ,  $C_{last}$ ,  $T_{last}$ ,  $C_{tau}$ ,  $AUC_{tau}$ , and T1/2 will be estimated.

For subjects in Part B, a single PK blood sample will be collected at all visits while on treatment for all subjects. The PK of SOF, GS-566500 and GS-331007 and/or ribavirin will be assessed.

The effect of age and SOF dose on PK (SOF and GS-331007) will be explored.

### **Statistical Methods:**

For Part A, plasma PK parameters  $C_{max}$ ,  $T_{max}$ ,  $C_{last}$ ,  $T_{last}$ ,  $C_{tau}AUC_{tau}$ , and  $T_{1/2}$  will be estimated. The PK parameters will be summarized by cohort. The effect of age and SOF dose on PK (SOF and GS-331007) will be explored.

For Part B, the primary efficacy endpoint is SVR12 in all enrolled and treated subjects. Secondary endpoints are SVR4, SVR24, breakthrough and relapse. Efficacy endpoints will be summarized by age group and genotype. Point estimate and its 95% confidence interval will be provided.

Subgroup analysis on SVR24 and SVR12 will be performed by treatment experience (treatment-naive vs. experienced) and by treatment experience and genotype. Other clinically relevant subgroup analyses may be conducted as appropriate (i.e., assuming that adequate numbers of patients in these subsets are available for analysis).

All continuous endpoints will be summarized using an 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum All categorical endpoints will be summarized by number and percentage of subjects who meet the endpoint definition.

Safety endpoints will be analyzed by the number and percent of subjects with events or abnormalities for categorical values or 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data by treatment group.

With approximately 50 subjects enrolled into each age group of Part B, a two-sided 95.0% confidence interval of the SVR12 rate will extend at most 11.1% in both directions from the observed SVR12 rate, assuming the expected SVR24 rate is 80%.

This study will be conducted in accordance with the guidelines of Good Clinical Practices (GCPs) including archiving of essential documents.

### GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS

° C degrees Celsius
° F degrees Fahrenheit

β-hCG β-human chorionic gonadotropin

AE adverse event

ALT alanine aminotransferase (also SGPT)

ANC absolute neutrophil count

APTT activated partial thromboplastin time
AST aspartate aminotransferase (also SGOT)

AUC area under the curve

AUC<sub>tau</sub> area under the plasma concentration versus time curve over the dosing

interval (tau)

BID twice a day

BLQ below the lower limit of quantification

BMI body mass index BW body weight

CL<sub>cr</sub> creatinine clearance

 $C_{max} \hspace{1.5cm} \hbox{the maximum observed serum/plasma/peripheral blood mononuclear} \\$ 

(PBMC) concentration of drug

C<sub>tau</sub> observed drug concentration at the end of the dosing interval (tau)

CMH Cochran-Mantel-Haenszel

COPD Chronic obstructive pulmonary disease

CRF case report form(s)

CRO Contract (or clinical) research organization

DAA Direct acting antiviral

dL Deciliter

DNA deoxyribonucleic acid

DMC Data Monitoring Committee

DSPH Drug Safety and Public Health

ECG Electrocardiogram

eCRF Electronic case report form(s)
ESA Erythropoiesis stimulating agent

Emax maximal effect
EU European Union

EVR Early virologic response

FAS full analysis set

FDA (United States) Food and Drug Administration
FEV<sub>1</sub> forced expiratory volume in one second
GCP Good Clinical Practice (Guidelines)
GCSF Granulocyte colony stimulating factor

# GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS (CONTINUED)

GGT gamma glutamyl transferase

 $\begin{array}{lll} \text{GSI} & \text{Gilead Sciences, Inc.} \\ \text{GT} & \text{Genotype (viral)} \\ \text{Hb} & \text{Hemoglobin} \\ \text{HbA}_{1c} & \text{Hemoglobin A}_{1c} \\ \text{HBV} & \text{Hepatitis B virus} \\ \text{HCV} & \text{Hepatitis C virus} \\ \end{array}$ 

HDPE high-density polyethylene

HIV Human Immunodeficiency Virus

HLGT High-Level Group Term

HLT High-Level Term

ICH International Conference on Harmonisation

IEC independent ethics committee

IL28B gene

IND Investigational New Drug (Application)

IRB institutional review board

IUD intrauterine device

IV Intravenous

IWRS interactive web response system

kg Kilogram L Liter

LDH Lactase dehydrogenase

LLN lower limit of the normal range

LLOD Lower limit of detection
LLOQ Lower limit of quantification

LLT Lower-Level Term

MedDRA Medical Dictionary for Regulatory Activities

Mg Milligram

MH Mantel-Haenszel

mL Milliliter
Min Minute

mmHg millimeters mercury NS (3/4A/5A/5B) Non-structural Protein

PBMC peripheral blood mononuclear cell(s)

PEG peginterferon alfa-2a
P-gp P-glycoprotein
PI Protease inhibitor
PK Pharmacokinetic

# GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS (CONTINUED)

QD once daily (use only in tables)

QTcF QT interval corrected using Fridericia' formula

RBC Red blood cell count

RBV Ribavirin

RDRP RNA-dependent RNA polymerase

RNA ribonucleic acid

RVR rapid virologic response
SADR Serious adverse drug reaction

SAE serious adverse event
SD Standard deviation
SOC Standard of Care

SOP Standard operating procedure

SUSAR Suspected Unexpected Serious Adverse Reaction

SVR Sustained Virologic Response

tmax The time (observed time point) of Cmax

TND Target not detected

TSH Thyroid stimulating hormone

t½ An estimate of the terminal elimination half-life of the drug in

serum/plasma/PBMC, calculated by dividing the natural log of 2 by the

terminal elimination rate constant ( $\lambda z$ )

ULN upper limit of the normal range

US United States

WBC white blood cell count

# 1. INTRODUCTION

# 1.1. Background

Hepatitis C virus (HCV) is responsible for a large proportion of chronic liver disease worldwide and accounts for 70% of cases of chronic hepatitis in industrialized countries. The global prevalence of chronic hepatitis C is estimated to average 3% {19705}.

The natural history of chronic HCV infection in children differs from that in adults since HCV infection in children is relatively benign. Most children chronically infected with HCV are asymptomatic or have mild nonspecific symptoms. Clinical symptoms are present in approximately 20% of children in the first 4 years of life, with hepatomegaly being the most frequent sign (10%). Many, but not all, perinatally infected children will have intermittently or persistently abnormal ALT or aspartate aminotransferase (AST) levels, particularly in the first 2 years of life. In children with vertical HCV infection who have undergone liver biopsy, the histological spectrum is usually mild, although severe liver disease is encountered {19801}. Despite the overall more favorable prognosis compared to adults, approximately 4% to 6% of children with chronic HCV infection have evidence of advanced fibrosis or cirrhosis and some children eventually require liver transplantation for end-stage liver disease as a consequence of HCV infection {19799}.

The goal of HCV treatment in both pediatric and adult populations is eradication of the virus, thereby preventing hepatic inflammation, hepatic fibrosis, cirrhosis, and liver failure resulting in either death or need for liver transplantation. This goal, however, is limited by the nature of the disease and the fact that not all patients are suitable candidates for currently approved treatments. In addition, pediatric treatment is controversial as the current treatment options are limited and severe side effects and tolerability can significantly limit or preclude their use. Despite well-established guidelines for the treatment of HCV in adults, there is no universal consensus on when or if to treat chronic HCV infection in children. In 2010, the European Society for Paediatric Gastroenterology, Hepatology, and Nutrition (ESPGHAN) issued guidance for clinical trial development for chronic HCV infection in children {20286}. In the guideline, the ESPGHAN suggested that the primary goal of treatment in children is to eradicate the infection to prevent late complications. Hence, the goal is not the treatment of an ongoing liver disease, but rather the prevention of a future one.

PEG and weight-based RBV are currently considered the standard of care for the treatment of HCV infection in children. Current recommendations are that patients with GT-2 or GT-3 be treated with PEG+RBV for 24 weeks and those with GT-1 or GT-4 should receive 48 weeks of therapy. Successful treatment of GT-1, however, has proved very difficult to achieve in spite of additional therapy or increased duration of treatment. A number of pediatric studies have reported that despite 48 weeks of treatment, sustained virologic response (SVR24) was observed in only 36% to 53% of subjects with GT-1, while response rates were > 80% in subjects with GT-2 or GT-3 {20285}.

Most children treated with PEG+RBV experience at least 1 adverse event due to treatment {20285}. Although most of these events are mild to moderate in severity, many of them result in dose reductions of 1 or both of the drugs. The most common adverse events have consisted of influenza-like illness (91%), headache (62%), and injection site reactions (45%), often leading to poor compliance and/or discontinuation from treatment.

Additionally, the concern for growth and development in this age group and the role that both PEG and RBV potentially play in reducing growth rates has initiated significant debate among pediatric hepatologists as to whether these treatments should even be considered in the pediatric population {20282}. Many pediatricians currently advocate delay of treatment past adolescence or even into adulthood when options with DAAs are possible {20282}. Unfortunately, in the 25% of pediatric patients who do meet the criteria for treatment (elevated transaminases and viral loads), the option of PEG+RBV therapy remains inadequate in regard to both efficacy in GT-1 and safety due to the many risks associated with this treatment.

Novel anti-hepatitis C treatments under study are directed against a variety of molecular targets, which include the virally encoded RNA-dependent RNA polymerase (RDRP, NS5B) and proteases (NS2 and NS3). Some of the most consistently effective antivirals have been nucleoside/tide analogs. These compounds share characteristics with the natural nucleoside substrates found in the cell, and once phosphorylated to the nucleoside-triphosphate, cause termination of the newly encoded viral genome.

SOF is a novel nucleotide analogue that inhibits HCV RNA replication in vitro and has demonstrated efficient inhibition of viral replication in in vitro and in vivo studies.. Furthermore, even in subjects who did experience off-treatment viral breakthrough, population sequencing revealed no treatment-emergent S282T mutations. No adverse effects on the nervous, cardiovascular, or respiratory systems have been observed, and no specific target organs of toxicity have been identified in long-term toxicology studies. Available clinical data indicate SOF has a favorable safety profile and is well tolerated.

Based on its observed safety and efficacy in adult patients with HCV, SOF has the potential to be a safe, tolerable, and effective treatment for HCV infection in the pediatric population.

### 1.2. Sofosbuyir

Sovaldi<sup>™</sup> (Sofosbuvir) is a potent nucleotide analogue that inhibits HCV RNA replication in vitro and has demonstrated high rates of sustained viral response (SVR) when given with RBV +/- PEG to subjects with chronic GT- 1, 2, 3 or 4 HCV infection {27503}, {23275}, {24713}, {24715}. Sovaldi has been approved in the United States by the Food and Drug Administration (FDA) for the treatment of HCV infection GT- 1, 2, 3 and 4 including treatment naïve and experienced patients and HIV/HCV co-infected patients.

For further information on the clinical pharmacology, virology, safety and efficacy of SOF, please refer to the current version of the Investigator's Brochure and US prescribing information.

# 1.3. Ribavirin (RBV)

Ribavirin is a guanosine analogue that inhibits the in vitro replication of a wide range of RNA and DNA viruses {15572}, {15668}. Ribavirin monotherapy has little or no effect on the replication of HCV but can result in normalization of serum ALT activity and improvement in liver histology. When combined with interferon or PEG therapy, RBV decreases substantially the relapse rate seen after cessation of interferon therapy {12557}, {12558}.

Ribavirin is a known teratogen (FDA category X). Furthermore, RBV is known to accumulate intracellularly where it is cleared slowly, and is also excreted in semen. Therefore, extreme care must be taken to avoid pregnancy during RBV therapy and for up to 7 months following completion of treatment. A comprehensive review of RBV is contained in the package insert/SmPC.

# 1.4. Rationale for the Current Study

This clinical study is designed to evaluate the efficacy and safety of treatment with SOF+RBV for adolescents and children with GT-2 and GT-3 chronic HCV infection.

Currently PEG and weight-based RBV are considered the standard of care for the treatment of HCV infection in children. However, this PEG and RBV regimen is long in duration, relatively toxic, and not well tolerated. Thus, there continues to be a need for new treatments for HCV that combine potent and sustained efficacy with improved tolerability and safety. Therapy that provides shorter duration and improved efficacy with an all-oral regimen would be a significant advancement over current options in pediatric patients.

The main aim for the treatment of pediatric patients with HCV is to eliminate the need to use IFN-based regimens. In this way, pediatric patients are able to avoid the necessity of weekly injections, which can be traumatic and burdensome, and also to significantly reduce the serious adverse events seen on administration of IFN-based regimens.

SOF is a promising candidate to combine with RBV based on its acceptable safety profile and its antiviral activity. Clinical trials from adult studies have demonstrated the antiviral efficacy, potency, and safety of SOF in subjects with HCV infection. SOF in combination with RBV would provide an all-oral, IFN-free regimen with a shorter treatment duration (12 - 24 weeks of SOF treatment versus standard-of-care 24 to 48 weeks of treatment) and would offer another important option in the treatment of HCV infection in the pediatric population.

While emerging Phase 3 data demonstrate high SVR12 rates in subjects with GT- 2 HCV infection, these studies suggest that patients with GT- 3 infection may benefit from a longer treatment duration with SOF+RBV. Optimal duration of SOF+RBV, for genotype 3 subjects, was established in FISSION and VALENCE. Increasing treatment duration from 12 to 24 weeks increased SVR12 from 61 to 93% in non-cirrhotics and from 34 to 92% in cirrhotics

### 1.5. Rationale for Dose Selection of SOF

SOF 400 mg, once daily, when dosed in combination with RBV with or without PEG has demonstrated broad genotypic efficacy and favorable safety profile in over 3300 HCV-infected subjects across multiple patient populations in Phase 2 and 3 trials. This dose is the marketed dose of SOF for the treatment of HCV-infection.

Selection of doses of SOF for adolescents and younger age groups will target systemic exposures similar to those observed in adults at the marketed dose, taking into account body weight/body surface area, the potential ontogenic changes in hepatically expressed carboxylesterase 1 (CES1) and Cathepsin A (CatA) enzymes, and the results obtained in older age groups. Available data suggest comparable hepatic expression of CES1 in adolescents and adults, with modestly decreased expression in children. As such, the adult clinical dose, 400mg, will be evaluated in adolescents {20288}. Safety and PK data in the adolescent group (Cohort 1) in Part A, will inform dose selection for the younger age groups in addition to body weight/body surface area.

Age-appropriate formulations of SOF that offer an important option in the treatment of HCV infection in the pediatric population are planned for evaluation in children below 6 years of age or children who are unable to swallow a solid-dose formulation.

### 1.6. Overall Risk/Benefit Assessment

Although the majority of pediatric patients infected with HCV exhibit minimal hepatic sequelae despite active viral replication and inflammation, a subset of children and adolescents will require treatment. Studies suggest that 3 major categories of disease can occur within 10 years after putative HCV exposure: (1) undetectable viremia and normal ALT, (2) persistent yet uncomplicated mild liver disease, and (3) progression to end-stage liver disease {20273}. It is the last two groups of children in whom therapy may be indicated to prevent end-stage disease, either during childhood/adolescence or in early adulthood.

Given that the current standard of care for the treatment of children infected with HCV is PEG and RBV and these regimens are long in duration, relatively toxic, and not well tolerated, there continues to be a need for new treatments for HCV that combine potent and sustained efficacy with improved tolerability and safety.

SOF has demonstrated efficient inhibition of viral replication in in vitro and in vivo studies. Available clinical data indicate SOF has a favorable safety profile and is well tolerated. SOF in combination with RBV is likely to provide significant therapeutic benefit in the treatment of HCV infection in pediatric patients compared to currently available therapies in the following areas:

- Expected improved efficacy in a pediatric population compared to the current standard of care
- Expected improvement in safety and tolerability in relation to either adverse reactions or potential medication errors in the pediatric population compared to the current standard of care

- Improved dosing scheme or method of administration (oral compared to subcutaneously administration and reduced treatment duration) leading to improved safety, efficacy, tolerability, and compliance
- Expected availability of a clinically relevant age-appropriate formulation
- Different mechanism of action with potential advantage for the pediatric population in terms of improved efficacy and safety
- Expected improvement in quality of life (eg, minimized duration of therapy and avoidance of IFN-related adverse events that affect patient quality of life such as flulike syndrome and depression)

Additionally, the study sponsor will perform an ongoing review of safety data during the conduct of the study.

# 2. OBJECTIVES

The primary objective of Part A of this study is:

 To evaluate the steady state pharmacokinetics (PK) and confirm the dose of SOF in HCV-infected pediatric subjects

The secondary objective of Part A of this study is:

 To evaluate the safety and tolerability of 7 days of dosing of SOF in HCV-infected pediatric subjects

The primary objectives of Part B of this study are:

 To evaluate the safety and tolerability of SOF + ribavirin (RBV) for 12 or 24 weeks in HCV infected pediatric subjects with GT- 2 or 3, respectively

To determine the antiviral efficacy of SOF+RBV treatment in GT- 2 and GT- 3 HCV-infected subjects separately, as assessed by the proportion of subjects with SVR 12 weeks after completion of treatment (SVR12)

The secondary objectives of Part B of this study are:

- To determine the antiviral efficacy of SOF+RBV treatment in genotype 2 and genotype 3 HCV-infected subjects separately, as assessed by the proportion of subjects with SVR 4 and 24 weeks after completion of treatment (SVR4 and SVR24)
- To evaluate the kinetics of circulating HCV RNA during treatment and after completion of treatment
- To evaluate the emergence of viral resistance to SOF during treatment and after completion of treatment

The exploratory objective of this study is:



# 3. STUDY DESIGN

# 3.1. Treatment Plan and Regimen

This is an open-label, multi-cohort, two-part study evaluating the PK, safety, and antiviral activity of SOF in chronic HCV-infected pediatric subjects.

### 3.1.1. Part A

Part A (PK lead-in) will evaluate and/or confirm age appropriate SOF doses by analyzing PK, safety, and antiviral activity of SOF through 7 days of dosing for each cohort. Children aged 3 to < 6 years, children aged 6 to < 12 years and adolescents aged 12 to < 18 years with genotype (GT) 2 or 3 HCV infection and evidence of HCV RNA > 1000 IU/mL at study entry will be evaluated. Three cohorts of up to 10 subjects each will be sequentially enrolled:

- Cohort 1: 12 to < 18 years old weighing  $\le$  45kg
- <u>Cohort 2:</u> 6 to < 12 years old
- Cohort 3: 3 to < 6 years old

The study will start with Cohort 1. Subjects will receive SOF (400-mg adult tablet or  $4 \times 100$ -mg tablets if determined necessary based on SOF swallowability assessment) for 7 days with intensive PK conducted on Day 7. A SOF swallowability assessment will be administered on Day 1 in which subjects will be observed taking the first 400-mg SOF tablet to confirm the swallowability of the 400-mg tablet size in adolescents aged 12 to < 18 years. If, at Day 1 or any time during the study, a subject is unable to continue with the 400-mg tablet size he/she will be re-assigned to  $4 \times 100$ mg SOF tablets.

Following completion of study treatment in Cohort 1 (Part A) and pending PK and safety results from Cohort 1 (Part A), Cohort 2 will initiate and receive study treatment (age appropriate formulation). Following completion of study treatment in Cohort 2 (Part A) and pending PK and safety results from Cohort 2 (Part A), Cohort 3 will receive study treatment (age-appropriate formulation).

Subjects in each cohort (Cohorts 1, 2 and 3) will immediately enroll in Part B as they complete Day 7 of Part A. On completion of Day 7 of Part A; subjects (aged 3 to < 18 years) will immediately enroll in Part B. They will begin dosing with SOF + RBV with no interruption of study drug administration.

### 3.1.2. Part B

Part B will be initiated by cohort after confirmation of age-appropriate SOF dosage levels. Subjects who participated in Part A will immediately rollover into Part B (Day 1), with no interruption of study drug administration:

Children aged 3 to < 12 years (Group 2) and adolescents aged 12 to < 18 years (Group 1) with GT-2 or GT-3 infection and evidence of HCV RNA > 1000 IU/mL at study entry (those who were dosed in Part A will have met this criteria prior to enrollment) will be evaluated.

Subjects enrolled in Part B will receive the following regimen.

- GT-2 subjects: SOF + RBV for 12 weeks
- GT-3 subjects: SOF + RBV for 24 weeks

The study will enroll both treatment-naïve and treatment-experienced pediatric subjects, with up to 20 subjects allowed to be treatment experienced. Approximately 100 total subjects, including subjects from Part A, will be enrolled in Part B as follows:

- Group 1: Approximately 50 adolescent subjects (12 to < 18 years of age)
- Group 2:Approximately 50 pediatric subjects (3 to < 12 years of age)

The following definitions will be used for treatment-experienced subjects:

- <u>Interferon intolerant:</u> Subject who discontinued therapy (≤ 12 weeks total) due to > 1 adverse event
- <u>Interferon non-responder:</u> Subject who did not achieve undetectable HCV RNA levels while on treatment
- Relapse/breakthrough: Subject who achieved undetectable HCV RNA during treatment or within 4 weeks of the end of treatment but did not achieve a sustained virologic response (SVR)

All subjects who do not attain SVR or have viral relapse will be encouraged to discuss treatment with standard-of-care (SOC) therapy with their healthcare provider.

Figure 3-1. Study Schema



# 3.2. Visit Schedule

### 3.2.1. Part A

Screening assessments will be completed within 28 days of the Day 1 visit.

Study Visits will occur at Screening, Day 1, Day 3, and Day 7.

Subjects (up to 10 subjects) enrolled in Part A will participate in an intensive PK evaluation on Day 7.

Following completion of the Day 7 intensive PK visit, subjects will then return for scheduled study visits outlined in Part B and begin dosing with SOF + RBV with no interruption of study drug administration.

### 3.2.2. Part B

Screening assessments will be completed within 28 days of the Day 1 visit. For subjects continuing from Part A, screening for Part B will not be required.

- **GT-2 Subjects:** Study visits for GT-2 subjects will occur at screening, Day 1, and the end of weeks 1, 2, 4, 8, and 12.
- **GT-3 Subjects:** Study visits for GT-3 subjects will occur at screening, Day 1, and the end of weeks 1, 2, 4, 8, 12, 16, 20, and 24.

All Part B subjects will then return for follow-up visits at 4, 12 and 24 weeks after discontinuation of therapy.

The total time to complete all study visits is approximately 40 or 52 weeks including:

- 28 day (4 week) screening period
- 12 or 24 week treatment period
- 24 week post-treatment period

The assessments performed at each visit are described in Section 6.

### 3.3. Virologic Response-Based Stopping Criteria

HCV RNA will be unblinded to the Investigator and Sponsor.

The following on-treatment virologic response-based treatment stopping criteria will be utilized:

- Confirmed HCV RNA ≥LLOQ after 2 consecutive HCV RNA <LLOQ
- Confirmed >1 log<sub>10</sub> increase from nadir
- HCV RNA ≥LLOQ through 8 weeks of treatment

Confirmation should be performed as soon as possible but within 2 weeks after determination of initial observation.

### 3.4. Treatment Discontinuations Criteria

The Medical Monitor should be consulted prior to subject discontinuation when medically feasible. Study medication must be discontinued in the following instances:

- Unacceptable toxicity, as defined in Section 7 of the protocol, or toxicity that, in the
  judgment of the investigator, compromises the ability to continue study-specific
  procedures or is considered to not be in the subject's best interest.
- Pregnancy of female subject or female partner of male subject.
- Efficacy failure as defined in Section 3.3.
- Significant protocol violation including non-compliance with study assessments.
- Subject request to discontinue for any reason; it is important to determine whether the withdrawal of consent is primarily due to an AE, lack of efficacy or other reason.
- Discontinuation of the study at the request of Gilead, regulatory agency or an Institutional Review Board (IRB)/Independent Ethics Committee (IEC).

### 3.5. Discontinuations

Subjects discontinuing treatment prior to completion of the assigned dosing period should complete an Early Termination visit as described in the Section 6.4.7.

Subjects who permanently discontinue all study drugs for any reason including safety and/or tolerability concerns prior to completion of the assigned dosing period will be followed according to the post-treatment study assessments described in Section 6.5.

# 3.6. Pharmacogenomic Substudy



# 3.7. Long Term Follow Up

All subjects (those who attain SVR24 or those who do not attain SVR24) who do not initiate other experimental or approved anti-HCV therapy will be followed every 6 months for assessments of growth, quality of life, and long-term viral suppression (if applicable) in a separate protocol. This follow-up will continue for 5 years. SUBJECT POPULATION

# 4. SUBJECT POPULATION

# 4.1. Number of Subjects and Subject Selection

Approximately 100 subjects will be enrolled in this study.

In order to manage the total study enrollment, Gilead Sciences, Inc., at its sole discretion, may suspend screening and/or discontinue the enrollment at any site at any time (upon written notice to the site). Discontinuation of the enrollment phase may result in the immediate ineligibility of all subjects screened but not yet enrolled, regardless of the progress or outcome of the screening assessments performed.

# 4.2. Inclusion Criteria

Subjects must meet *all* of the following inclusion criteria to be eligible for participation in this study.

- 1. Parent or legal guardian able to provide written informed consent prior to any screening evaluations and willing to comply with study requirements
- 2. 3 years to < 18 years of age (consent of parent or legal guardian required)
- 3. Part A only: subjects in Cohort 1 (age 12 to <18 years of age) must weigh  $\ge$  45 kg
- 4. Documented chronic HCV infection, GT-2 or GT-3
- 5. HCV RNA ≥ 1000 IU/mL at Screening
- 6. Adequate hematologic function (absolute neutrophil count  $\geq$  1,500/mm<sup>3</sup>; hemoglobin  $\geq$  10.0 g/dL)
- 7. Negative serum β-HCG pregnancy test (for females of childbearing potential only, as defined in Appendix 5)
- 8. Subject able to provide written assent, if they have the ability to read and write, as determined by IRB/IEC/local requirements and Investigator's discretion

### 4.3. Exclusion Criteria

Subjects who meet *any* of the following exclusion criteria are not to be enrolled in this study.

- 1. Pregnant or lactating subjects
- 2. Sexually-active males or females of childbearing potential who are not willing to use an effective method of contraception during the study (see Appendix 5 for further details)

- 3. Decompensated liver disease defined as INR > 1.2 × ULN, platelets < 50,000/mm<sup>3</sup>, serum albumin < 3.5 g/dL, or prior history of clinical hepatic decompensation (e.g., ascites, jaundice, encephalopathy, variceal hemorrhage)
- 4. Chronic liver disease of a non-HCV etiology (eg, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency)
- 5.  $\alpha$ -fetoprotein > 50 ng/mL
- 6. Serum creatinine > 1.5 mg/dL
- 7. Evidence of hepatocellular carcinoma (HCC)
- 8. Co-infection with HIV, acute HAV, or HBV
- 9. Significant cardiovascular, pulmonary or neurological disease
- 10. Evidence of a gastrointestinal malabsorption syndrome that may interfere with absorption of orally administered medications
- 11. History of solid organ or bone marrow transplantation
- 12. Chronic daily non-steroidal anti-inflammatory drug therapy
- 13. Systemic corticosteroid use for  $\geq 5$  days (pulmonary/nasal administration is permitted)
- 14. Investigational agents (except with the expressed approval of the Sponsor)
- 15. Clinically-relevant alcohol or drug abuse within 12 months of screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by the investigator
- 16. Known hypersensitivity to the study drugs, the metabolites or formulation excipients
- 17. Any other condition (including alcohol or substance abuse) or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements
- 18. Use of any prohibited concomitant medications as described in Section 5.6 within 28 days of the Day 1 visit

# 5. INVESTIGATIONAL MEDICINAL PRODUCTS

# 5.1. Randomization and Blinding

Not applicable.

### 5.2. Sofosbuvir

# 5.2.1. Description and Handling

### 5.2.1.1. Formulation:

SOF tablets, 400 mg, are yellow, capsule-shaped, film-coated tablets debossed with "GSI" on one side and "7977" on the other side. In addition to the active ingredient, SOF tablets contain the following inactive ingredients: mannitol, microcrystalline cellulose, croscarmellose sodium, colloidal silicon dioxide, magnesium stearate, polyvinyl alcohol, titanium dioxide, macrogol, talc, and yellow iron oxide.

SOF tablets, 100 mg, are yellow, round, film-coated, plain-faced tablets. In addition to the active ingredient, SOF tablets contain the following inactive ingredients: mannitol, microcrystalline cellulose, croscarmellose sodium, colloidal silicon dioxide, magnesium stearate, polyvinyl alcohol, titanium dioxide, macrogol, talc, and yellow iron oxide.

Ages appropriate formulations for children aged 3 to < 12 years are to be determined.

# 5.2.1.2. Packaging and Labeling

SOF 400 mg tablets are packaged in white, high density polyethylene (HDPE) bottles. Each bottle contains 30 tablets and a silica gel desiccant canister or sachet and polyester packing material. Each bottle is enclosed with a white, continuous thread, child-resistant screw cap with an induction-sealed, aluminum-faced liner.

SOF 100 mg tablets are packaged in white, high density polyethylene (HDPE) bottles. Each bottle contains 28 tablets and a polyester packing material. Each bottle is enclosed with a white, continuous thread, child-resistant screw cap with an induction-sealed, aluminum faced liner.

SOF bottles to be distributed to centers in the US, EU and the rest of the countries will meet all applicable requirements of the US Food and Drug Administration (FDA) and Annex 13 of Good Manufacturing Practices: Manufacture of investigational medicinal products (July 2010) and/or other local regulations as applicable.

### 5.2.2. Storage and Handling

SOF tablets should be stored at controlled room temperature until required for administration. Controlled room temperature is defined as 25 °C (77 °F); excursions are permitted between 15 °C and 30 °C (59 °F to 86 °F).

All drug products should be stored in a securely locked area, accessible only to authorized site personnel. To ensure the stability of the study drug and to ensure proper product identification, the drug product should not be stored in a container other than the container in which they are supplied. Consideration should be given to handling, preparation, and disposal through measures that minimize drug contact with the body. Appropriate precautions should be followed to avoid direct eye contact or exposure through inhalation when handling SOF.

Sufficient quantities of SOF tablets to complete the entire study will be shipped to the investigator or qualified designee from Gilead Sciences Materials & Logistics (or its designee).

# **5.2.3.** Dosage and Administration of SOF

### Age group 12 to < 18 years:

Part A: SOF 400-mg tablets will be administered once daily. Subjects determined unable to swallow the 400-mg tablet, by SOF swallowability assessment at Day 1 or any time during the study, will be re-assigned to 4 x 100-mg tablets daily.

Part B: SOF 400-mg tablets will be administered once daily for subjects who weigh  $\geq$  45 kg. Subjects determined unable to swallow the 400-mg tablet (by SOF assessment at Day 1 or at any time during the study) will be re-assigned to 4 x 100-mg tablets daily. For subjects in this age group who weigh < 45 kg, PK data from part A will be used to determine the appropriate dose of SOF to be administered.

Subjects who participated in Part A will continue the assigned dose in Part B.

### Age group 3 to < 12 years:

SOF age-appropriate formulation will be administered once daily with a dose and formulation to be determined.

### 5.3. Ribavirin

# **5.3.1.** Description and Handling of RBV

### 5.3.1.1. Formulation

RBV tablets, 200 mg, are blue, capsule-shaped, film-coated tablets debossed with "3RP" on one side and "200" on the other side. In addition to the active ingredient, RBV tablets contain the following inactive ingredients: microcrystalline cellulose, lactose monohydrate, croscarmellose sodium, povidone, magnesium stearate, polyvinyl alcohol), titanium dioxide, macrogol, talc and FD&C blue #2.

RBV Oral Solution 40 mg per mL is a clear, colorless to pale or light yellow bubble gum-flavored liquid. In addition to the active ingredient, RBV oral solution contains the following inactive ingredients: sucrose, glycerin, sorbitol, propylene glycol, sodium citrate, citric acid, sodium benzoate, natural and artificial flavor for bubble gum #15864, and water.

### 5.3.1.2. Packaging and Labeling

The RBV tablets are packaged in white, HDPE bottles. Each bottle contains 168 tablets and rayon coil packing material and is enclosed with a white, continuous thread, child-resistant screw cap with an induction-sealed, aluminum-faced liner.

The RBV oral solution is packaged in 4-oz amber glass bottles (100 mL/bottle) with child-resistant closures.

RBV bottles to be distributed to centers in the US, EU and the rest of the countries will meet all applicable requirements of the US Food and Drug Administration (FDA) and Annex 13 of Good Manufacturing Practices: Manufacture of investigational medicinal products (July 2010) and/or other local regulations as applicable.

# 5.3.1.3. Storage and Handling

RBV tablets should be stored at 25 °C (77 °F); excursions are permitted between 15 and 30 °C (59 and 86 °F).

RBV oral solution should be stored between 2-8°C (36-46°F) or at 25°C (77°F); excursions permitted to 15-30°C (59-86°F).

### **5.3.2.** Dosage and Administration of RBV

RBV dose will be administered by weight as follows:

- Below 50 kg: RBV 15 mg/kg divided BID
- 50 kg to < 65 kg : RBV 400 mg BID
- 65 kg to < 75 kg: RBV 400 mg in the morning and 600 mg in the evening
- Greater than or equal to 75 kg: 600 mg BID

The morning dose of RBV will be taken with SOF and food. The evening dose of RBV will be taken with food.

RBV tablets will be supplied by Gilead Sciences for all subjects.

### 5.4. Co-administration of SOF and RBV

In Part B of the study, each subject will be given instructions to maintain approximately the same daily dosing interval between study drug doses.

For **morning doses**, subjects will be instructed to take study drugs with food as follows:

- SOF
- Weight-based RBV (as per Section 5.3.2).

For <u>evening doses</u>, subjects will be instructed to take study drug with food as follows:

• Weight-based RBV (as per Section 5.3.2).

If a subject forgets to take the medication at the correct time, it may be taken later in the day; however, no more than 400 mg dose of SOF should be taken on any calendar day. The subject should resume the standing dosing schedule on the next day. Study medications should not be cut or split.

# 5.5. Study Drug Compliance

Subjects will be instructed to return any unused SOF and RBV in the original container on Day 7 (Part A) and/or at study treatment visits every 4 weeks (Part B).

Returned medication will be reconciled by the investigator in order to monitor the subject's compliance with the medication regimen.

### **5.6.** Prior and Concomitant Medications

Concomitant medications taken within 30 days of Screening, up to and including the date of the visit four weeks after discontinuation of study treatment, need to be recorded in the source documents and eCRFs. All concomitant medications should be recorded in the source documents.

The following medications are prohibited from 28 days prior to the Day 1 visit through the end of treatment:

- Erythropoiesis-stimulating agents (ESAs); including but not limited to Procrit<sup>®</sup>, Aranesp<sup>®</sup> and Epogen<sup>®</sup>
- Granulocyte colony stimulating factor (GCSF)
- Chronic systemic immunosuppressants including corticosteroids (prednisone equivalent of > 10 mg/day for > 2 weeks), azathioprine, or monoclonal antibodies (e.g., infliximab)
- Investigational agents or devices for any indication
- Drugs disallowed per prescribing information of REBETOL<sup>®</sup>
- Concomitant use of certain medications or herbal/natural supplements (inducers of drug transporters i.e. P-gp) with study drug(s) may result in pharmacokinetic interactions resulting in decreases in exposure of study drug(s). Representative medications which are excluded from 21 days prior to Day 1 through the end of treatment are listed below:

| Drug | Agents Disallowed | Concomitant use with study drug may potentially result in changes of study drug concentration as listed below |
|---|---|---|
| Anticonvulsants | Phenobarbital, Phenytoin,<br>Carbamazepine, Oxcarbazepine | Decrease in concentration of study drug |
| Antimycobacterials | Rifampin, rifabutine, rifapentine | Decrease in concentration of study drug |
| Herbal/Natural<br>Supplements | St. John's Wort, Echinacea, Milk thistle (i.e., silymarin), Chinese herb sho-saikoto (or Xiao-Shai-Hu-Tang) | Decrease in concentration of study drug |

Medications for disease conditions **excluded** from the protocol (e.g., HIV-1 infection, active cancer, transplantation) are not listed under this Concomitant Medication section and are disallowed in the study.

# 6. STUDY PROCEDURES

All subjects will complete screening, on-treatment and post-treatment assessments. Screening assessments will be completed within 28 days of the Day 1 visit. The end of study will occur at the 24-week Post-Treatment visit. The schedule of assessments is described below.

Information on the specific laboratory parameters to be measured and clinical assessments to be performed are provided in Section 6.6.

# 6.1. Subject Enrollment

Each candidate's parent or legal guardian must sign an Informed Consent Form prior to the conduct of any screening procedures. Each study candidate who has the ability to read and write must sign an Assent Form, as required by IRB/IEC/local requirements, prior to the conduct of any study procedures. Screening evaluations will be used to determine the eligibility of each candidate for study enrollment. Candidates who fail to meet eligibility criteria by screening evaluations may be re-screened once  $\geq 30$  days after the initial screen if there is a reasonable expectation that the candidate will be eligible after repeat screening.

# **6.2.** Screening Assessments

# 6.2.1. Screening Visit (Day –28 to Day 0)

Subjects will complete all screening assessments within 28 days of the Day 1 visit. The screening window can be extended to 42 days for subjects requiring additional HCV genotype testing or for extenuating circumstances.

Subjects who participated in Part A will not require an additional screening visit prior to starting Part B.

The following procedures will be performed and documented:

- Written informed consent from parent or legal guardian and assent from subject, if applicable (see above)
- Medical history, including:
  - Hepatitis C history
  - Hepatitis C treatment history
  - Family history (i.e., height and weight of parents, if known)
  - Liver biopsy results within 2 years of Screening (if available)
- Complete physical examination

- (Part A only) Perform Tanner Pubertal Stage assessment for subjects ≥ 6 years of age at the time of the visit, until Tanner Stage 5 has been reached. Date of first menses will be documented
- Vital signs (temperature, blood pressure, pulse, respiratory rate), body weight and height
- Obtain blood samples for tests as listed in Section 6.6.1:
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Determination of HCV viral genotype and subtype
  - HCV antibody, HIV 1/2 antibody, and HBs antigen, HAV antibody
  - HbA<sub>1c</sub>
  - TSH
  - IL28B
  - Serum β-hCG pregnancy test for females of childbearing potential only
  - Alpha fetoprotein (AFP)
  - Alpha-1 anti-trypsin (ATT)
- Obtain urine sample for:
  - Urinalysis
  - Urine Drug Screen
- Review of concomitant medications
- Review of all inclusion and exclusion criteria

Subjects meeting all of the inclusion criteria and none of the exclusion criteria will return to the clinic for the Day 1 visit assessments.
#### 6.3. Part A: Treatment Assessments

#### 6.3.1. **Day 1 Visit**

After confirmation of eligibility has been evaluated, the following tests and procedures must be completed prior to enrollment and dosing/dispensing on Day 1:

- Perform complete physical examination
- Vital signs, including body weight and height
- Assessment of AEs and concomitant medications
- Pregnancy prevention counseling including partner pregnancy prevention for male participants (Subjects 12 to < 18 years of age only)
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral sequencing (archive)
- Obtain urine samples for the following procedures:
  - Urinalysis
  - β-hCG pregnancy test for females of childbearing potential only

### 6.3.1.1. Drug Administration

- Dispense study drugs as directed by the IWRS
- Instruct the subject on the appropriate RBV dose after weight-based dosage is calculated using Day 1 weight
- Instruct the subject on the packaging, storage and administration of all study drugs
- Perform SOF swallowability assessment (for subjects administered SOF in tablet form only)
- Observe the subject taking the first dose of study drugs (with food) and record the time of first dose

#### 6.3.2. Day 3

The following procedures/assessments are to be completed on Day 3:

- Perform a symptom-directed physical examination as needed
- Vital signs, including body weight and height
- Assessment of AEs and concomitant medications
- Review medication compliance with subject and/or parent/guardian
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - HCV RNA
  - Viral sequencing (archive)

# 6.3.3. Day 7 – Intensive PK

The Day 7 Intensive PK visit should occur on the protocol-specified visit date based on the Day 1 visit. For the purposes of scheduling, the Day 7 Intensive PK visit may be performed within +3 days of the protocol-specified visit date (Subjects will continue daily dosing through the Intensive PK Visit).

Subjects should come in a fasted state for the Day 7 Intensive PK visit (i.e., no food or drink except water at least 8 hours prior to the Day 7 Intensive PK visit). Subjects and/or parents/guardians should be instructed that the Day 7 dose of SOF must **not** be taken until the evaluations listed below are completed.

If the subject has already dosed prior to the Day 7 clinic visit or is **not** in a fasted state, the Day 7 intensive PK assessments must not be completed. The subject and/or parents/guardians should be instructed to return in a fasted state within 3 days (Days 8, 9, or 10) for the intensive PK visit. Appropriate study drug re-dispensation must be performed in this case.

If dosing non-compliance is identified on or prior to the Day 7 visit, the Day 7 intensive PK assessments must not be completed. The subject and/or parents/guardians should be counseled regarding proper dosing and be scheduled to return for the Day 7 intensive PK visit no sooner than 3 days following compliant dosing and no later than Day 11 (i.e., return on Day 10 or Day 11). If dosing non-compliance is due to an AE, consultation with the Gilead Medical Monitor is required regarding the potential of rescheduling the Day 7 intensive PK visit.

In both scenarios described above, the subject and/or parents/guardians should be reminded not to take the SOF prior to arriving at the clinic on the day of the re-scheduled intensive PK visit. All Day 7 intensive PK assessments listed below should be completed when the subject returns.

The following evaluations are to be completed at the Day 7 Intensive PK visit:

- Perform a symptom-directed physical examination as needed
- Vital signs, including body weight and height
- Assessment of AEs and concomitant medications
- Perform study drug accountability
- Review medication compliance with subject and/or parent/guardian.
- Obtain urine samples for the following procedures:
  - Urinalysis
  - Urine pregnancy test (females of childbearing potential only). If the urine pregnancy test is positive, the Intensive PK sampling will not be completed. The positive result will be confirmed with a serum pregnancy test.
- Obtain blood samples for the following laboratory analyses:
  - Hematology
  - Chemistry
  - HCV RNA
  - Viral sequencing (archive)
- Perform intensive PK sampling:
  - Blood samples will be collected at 0 (predose, ≤ 30 minutes prior to dosing). After collection of the predose sample, subjects will be provided a standardized meal. Within 5 minutes after consuming the standardized meal, subjects will be dosed with SOF per dosing requirements.

- Post-dose blood samples will be collected as follows:
  - For Cohorts 1 and 2: 0.5, 1, 2, 3, 4, 8, and 12 hours post-dose (with predose also serving as t= 24).
  - For Cohort 3 only: 2, 4, 8, and 12 hours post-dose (with predose also serving as t = 24).
- Subjects will be restricted from food intake until after collection of the 4-hour post dose blood sample, except for subjects in Cohort 3. Please also refer to the PK manual for details about standardized meals and PK sample processing instructions.

After completing the Day 7 intensive PK visit subjects will then continue to the Day 1 visit in Part B described in Section 6.4.1

#### 6.4. Part B: Treatment Assessments

#### 6.4.1. Day 1 Visit

After confirmation of eligibility has been evaluated, the following tests and procedures must be completed prior to enrollment and dosing/dispensing on Day 1:

- Perform complete physical examination
- Vital signs, including body weight and height
- Review of AEs and concomitant medications
- Pregnancy prevention counseling including partner pregnancy prevention for male participants (Subjects 12 to < 18 years of age only) Obtain blood samples for:</li>

| _ | Hematology |
|---|----------------------------|
| _ | Chemistry |
| _ | Coagulation tests |
| | HCV RNA |
| _ | Viral sequencing (archive) |
| | PPD |

- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Subject completes quality of life survey: Subject is to review questionnaire with a parent/guardian and write/mark answers directly onto the questionnaire.

## 6.4.1.1. Drug Administration

- Dispense study drugs as directed by the IWRS
- Instruct the subject on the appropriate RBV dose after weight-based dosage is calculated using Day 1 weight
- Instruct the subject on the packaging, storage and administration of all study drugs
- Observe the subject taking the first dose of study drugs (with food) and record the time of first dose
- Perform SOF swallowability assessment (for subjects administered SOF in tablet form only)

# 6.4.2. Weeks 1 and 2 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at these visits:

- Vital signs, including body weight and height
- Perform symptom-directed physical examination
- Assessment of AEs and concomitant medications
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral sequencing (archive)
  - Single PK

#### 6.4.3. Weeks 4 and 8 (± 3 days)

- Vital signs, including body weight and height
- Perform symptom-directed physical examination
- Assessment of AEs and concomitant medications
- Obtain blood samples for
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral sequencing (archive)
  - Single PK
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Review medication compliance with subject and/or parent/guardian (subject should return all study drugs at these visits)
- Dispense study drugs as directed by the IWRS

### 6.4.4. Week 12 ( $\pm$ 3 days)

- Perform complete physical examination
- Tanner Staging Assessment
- Vital signs, including body weight and height
- Assess Rates of Growth (percentiles)
- Assessment of AEs and concomitant medications
- Pregnancy prevention counseling including partner pregnancy prevention for male participants (Subjects 12 to < 18 years of age only)

- Obtain blood samples for:
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral sequencing (archive)
  - TSH
  - Single PK
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Subject completes quality of life survey: Subject is to review questionnaire with a parent/guardian and write/mark answers directly onto the questionnaire. (GT-2 Subjects only)
- Review medication compliance with subject and/or parent/guardian.
- Dispense study drugs as directed by the IWRS (GT-3 Subjects Only)
- GT-2 Subjects should return all bottles and kits at the Week 12 Visit

#### 6.4.5. Week 16 and 20 ( $\pm$ 3 days) – GT-3 Subjects only

- Vital signs, including body weight and height
- Perform symptom-directed physical examination
- Assessment of AEs and concomitant medications
- Obtain blood samples for
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral sequencing (archive)
  - Single PK

- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Review medication compliance with subject and/or parent/guardian (subject should return all study drugs at these visits)
- Dispense study drugs as directed by the IWRS

### 6.4.6. Week $24(\pm 3 \text{ days}) - \text{GT-3 Subjects only}$

- Perform complete physical examination
- Tanner Staging Assessment
- Vital signs, including body weight and height
- Assess Rates of Growth (percentiles)
- Assessment of AEs and concomitant medications
- Pregnancy prevention counseling including partner pregnancy prevention for male participants (Subjects 12 to < 18 years of age only)
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral sequencing (archive)
  - TSH
  - Single PK
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Subject completes quality of life survey: Subject is to review questionnaire with a parent/guardian and write/mark answers directly onto the questionnaire

- Review medication compliance with subject and/or parent/guardian.
- GT-3 Subjects should return all bottles and kits at the Week 24 Visit

# 6.4.7. Unscheduled Visit/Early Termination Visit

A subject should attend an unscheduled visit if requested by the sponsor or the investigator. The assessments are at the investigator's discretion.

The Sponsor/CRO should be informed when a subject comes off treatment due to an adverse event. If a subject discontinues treatment then the assessments outlined below should be performed.

- Perform complete physical examination
- Tanner Pubertal Stage Assessment
- Vital signs, including body weight and height
- Assess Rates of Growth (percentiles)
- Assessment of AEs and concomitant medications
- Pregnancy prevention counseling including partner pregnancy prevention for male participants (Subjects 12 to < 18 years of age only)
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral sequencing (archive)
  - TSH
  - Single PK
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Subject completes quality of life survey: Subject is to review questionnaire with a parent/guardian and write/mark answers directly onto the questionnaire.

- Review medication compliance with subject and/or parent/guardian.
- Subjects should return all bottles and kits at the Early Termination Visit

All subjects should complete Post-Treatment assessments after early termination, as described in Section 6.5.

#### 6.5. Post-Treatment Assessments

#### 6.5.1. 4-Week Post-Treatment Visit (± 5 days)

- Vital signs, including body weight and height
- Perform symptom-directed physical examination
- Assessment of AEs and concomitant medications
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - HCV RNA
  - Viral sequencing (archive)
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Pregnancy prevention counseling including partner pregnancy prevention for male participants (Subjects 12 to < 18 years of age only)

Female subjects of childbearing potential should be provided with Urine Pregnancy Test-Kits, instructed on their use and requested to continue to self-monitor for pregnancy for 6-months after their last dose of RBV. If required by local regulations, additional pregnancy tests beyond 6 months may be added. The subject should be contacted every 4 weeks and asked to report results of the urine pregnancy tests. If a positive urine pregnancy test is reported, the subject should return to the clinic for a serum pregnancy test.

#### 6.5.2. 12-Week Post-Treatment Visit (± 5 days)

- Vital signs, including body weight and height
- Perform symptom-directed physical examination

- Perform Tanner Pubertal Stage assessment for subjects  $\geq 6$  years of age at the time of the visit, until Tanner Stage 5 has been reached. Date of first menses will be documented.
- Obtain blood samples for
  - Hematology
  - Chemistry
  - HCV RNA
  - Viral sequencing (archive)
- Obtain urine sample for:
  - β-hCG pregnancy test for females of childbearing potential only
- Pregnancy prevention counseling including partner pregnancy prevention for male participants (Subjects 12 to < 18 years of age only)
- Subject completes quality of life survey: Subject is to review questionnaire with a parent/guardian and write/mark answers directly onto the questionnaire

# 6.5.3. 24-Week Post-Treatment Visit (± 5 days)

- Vital signs, including body weight and height
- Perform symptom-directed physical examination
- Tanner Pubertal Stage Assessment & Rates of growth
- Obtain blood samples for
  - HCV RNA
  - Viral sequencing (archive)
- Obtain urine sample for β-hCG pregnancy test for females of childbearing potential only
- Subject completes quality of life survey: Subject is to review questionnaire with a parent/guardian and write/mark answers directly onto the questionnaire.
- Pregnancy prevention counseling including partner pregnancy prevention for male participants (Subjects 12 to < 18 years of age only)

### 6.6. Procedures and Specifications

#### 6.6.1. Clinical Laboratory Analytes

<u>Hematology:</u> Hematocrit, Hemoglobin (Hb), Platelet count, Red blood cell count (RBC), White blood cell count (WBC) with differential (absolute and percentage) including Lymphocytes, Monocytes, Neutrophils, Eosinophils, Basophils, Reticulocyte count and MCV.

Coagulation: INR, Prothrombin time (PT), Activated partial thromboplastin time (APTT)

<u>Chemistry</u> Alanine aminotransferase (ALT/SGPT), Aspartate aminotransferase (AST/SGOT), Albumin, Alkaline phosphatase, Creatinine, Total Bilirubin (reflex to Direct Bilirubin), Glucose, Lipase, Potassium, Sodium, Gamma-glutamyl transferase (GGT), alpha fetoprotein (AFP), alpha-1 anti-trypsin.

<u>Urinalysis:</u> Appearance, Blood, Color, Glucose, Leukocyte esterase, pH, Protein, Urobilinogen. Reflex to microscopic urinalysis if dipstick result is abnormal.

<u>Virological Tests</u>: Serologies for HCV, HBV and HIV. HCV RNA will be measured using the COBAS<sup>®</sup> AmpliPrep/COBAS<sup>®</sup> TaqMan<sup>®</sup> HCV Test, v2.0 for Use with the High Pure System. HCV genotype and subtype will be determined using the Siemens VERSANT<sup>®</sup> HCV Genotype INNO-LiPA 2.0 Assay. Gilead reserves the right to use alternate assays for HCV RNA and HCV genotype should the above assays become unavailable.

IL28B genotype will be determined by polymerase chain reaction (PCR) amplification of the SNP, rs12979860, with sequence specific forward and reverse primers and allele specific fluorescently labeled TaqMan<sup>®</sup> MGB probes. Gilead reserves the right to use alternate assays for IL28B determination should the above assay become unavailable.

<u>Pregnancy Tests</u>: Serum β-hCG, Urine β-hCG (if positive, requires immediate confirmation with Serum β-hCG)

Additional Tests: Hemoglobin A1c (HbA1c), TSH (reflex Free T4), Alfa fetoprotein (AFP), Alpha-1 anti-trypsin (AAT)

# 6.6.2. Medical History

Medical history including details regarding illnesses and allergies, date(s) of onset, and whether condition(s) is currently ongoing, and medication history will be collected on all subjects during screening.

## 6.6.3. Complete Physical Examination

A complete physical examination must include source documentation of general appearance, and the following body systems: Head, neck and thyroid; eyes, ears, nose, throat, mouth and tongue; chest (excluding breasts); respiratory; cardiovascular; lymph nodes, abdomen; skin, hair, nails; musculoskeletal; neurological.

#### 6.6.4. Tanner Pubertal Stage Assessment

The Tanner Stage scale is available in Appendix 4

#### 6.6.5. Vital Signs

Assessment of vital signs will include measurement of resting blood pressure, pulse, respiratory rate, and temperature.

Blood pressure will be measured using the following standardized process:

- Subject should sit for  $\geq 5$  minutes with feet flat on the floor and measurement arm supported so that the midpoint of the manometer cuff is at heart level;
- Use a mercury sphygmomanometer or automatic blood pressure device with an appropriately sized cuff with the bladder centered over the brachial artery;
- Measure and record the blood pressure to the nearest 2 mmHg mark on the manometer or to the nearest whole number on an automatic device.

## 6.6.6. Body Mass Index (BMI)

BMI is calculated by the following equation.

BMI = 
$$\underbrace{\text{weight (pounds)} \times 703}_{\text{(height in inches)}^2}$$
 or  $\underbrace{\text{weight in kilograms}}_{\text{(height in meters)}^2}$ 

# 6.6.7. Viral Sequencing (Archive)

Plasma samples will be collected at Day 1 and each visit for viral sequence analysis. Unused samples may be archived.

#### 6.6.8. Pregnancy Testing

All females of childbearing potential will have urine pregnancy testing every 4 weeks during the dosing period and for a minimum of 6 months following the last dose of RBV. If required by local regulations, additional pregnancy tests beyond 6 months may be added. In the event of a positive urine pregnancy result, subjects will be instructed to stop study drugs immediately and return to the clinic as soon as possible for a serum pregnancy test.

Pregnancy test kits will be dispensed to female subjects of child bearing potential at the 4-Week Post-Treatment visit. The subject will be contacted by telephone monthly to confirm that urine pregnancy testing has been performed post-treatment and to record the outcome.

Alternatively, if required by local regulations or preferred by the investigator or subject, the subject may return to the clinic for urine pregnancy tests.

# 6.6.9. Quality of Life Survey (PedsQL $^{\text{TM}}$ )

The survey will be completed in Part B of the study at Day 1, End of Treatment (Week 12 for GT-2 subjects, Week 24 for GT-3 subjects, or at Early Termination, if applicable), 12-Week Post-Treatment, and 24-Week Post-Treatment visits.

#### 7. TOXICITY MANAGEMENT

# 7.1. Modification of Dose/Schedule Due to Toxicity

#### 7.1.1. RBV Dose Adjustments

No formal RBV dose reduction guidelines exist for pediatric patients. Prior to RBV dose adjustments, the Gilead Medical Monitor should be consulted.

#### 7.2. Subject Stopping Rules for SOF

The Gilead Medical Monitor should be consulted prior to dose discontinuation of SOF unless the investigator believes that immediate action is warranted to ensure the continued safety of the subject.

Administration of SOF may be discontinued due to a clinical or laboratory event. There is no option for SOF dose reduction. If SOF is stopped for toxicity, it should not be restarted, RBV should be stopped and the subject should complete an Early Termination Visit.

Subjects who meet any of the following laboratory criteria should stop treatment with SOF and RBV:

- Elevation of ALT and/or AST >5x Day 1 or nadir, confirmed by immediate repeat testing
- Abnormal elevation of ALT >3x Day 1 and total bilirubin >2 x ULN, confirmed by immediate repeat testing
- Confirmed elevation of ALT >15 x ULN
- Any Grade 3 or greater rash associated with constitutional symptoms
- Any Grade 4 event or lab abnormality assessed as related to treatment with SOF

#### 8. ADVERSE EVENTS MANAGEMENT

# 8.1. Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events

#### 8.1.1. Adverse Events

An adverse event (AE) is any untoward medical occurrence in a clinical study subject administered a pharmaceutical product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs may also include pre- or post- treatment complications that occur as a result of protocol-mandated procedures, overdose, drug abuse/misuse reports, or occupational exposure. Preexisting events that increase in severity or change in nature during or as a consequence of participation in the clinical study will also be considered AEs.

An AE does not include the following:

- Medical or surgical procedures such as surgery, endoscopy, tooth extraction, and transfusion. The condition that led to the procedure may be an adverse event and must be reported
- Pre-existing diseases, conditions, or laboratory abnormalities present or detected before the screening visit that do not worsen.
- Situations where an untoward medical occurrence has not occurred (e.g., hospitalization for elective surgery, social and/or convenience admissions).
- Overdose without clinical sequelae (see Section 8.5)
- Any medical condition or clinically significant laboratory abnormality with an onset date before the consent form is signed and not related to a protocol-associated procedure is not an AE. It is considered to be pre-existing and should be documented on the medical history CRF

#### 8.1.2. Serious Adverse Events

A **serious adverse event** (SAE) is defined as an event that, at any dose, results in the following:

- Death
- Life-threatening (Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.)

- In-patient hospitalization or prolongation of existing hospitalization
- Persistent or significant disability/incapacity
- A congenital anomaly/birth defect
- A medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs. Medical and scientific judgment must be exercised to determine whether such an event is reportable under expedited reporting rules. Examples of medically important events include intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; and development of drug dependency or drug abuse. For the avoidance of doubt, infections resulting from contaminated medicinal product will be considered a medically important event and subject to expedited reporting requirements.

# 8.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events

Laboratory abnormalities without clinical significance are not recorded as AEs or SAEs. However, laboratory abnormalities (eg, clinical chemistry, hematology, and urinalysis) that require medical or surgical intervention or lead to IMP interruption, modification, or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (eg, electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE or SAE as described in Sections 8.1.1 and 8.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (eg, anemia), not the laboratory result (ie, decreased hemoglobin).

#### 8.2. Assessment of Adverse Events and Serious Adverse Events

The investigator or qualified subinvestigator is responsible for assessing AEs and SAEs for causality and severity, and for final review and confirmation of accuracy of event information and assessments.

### 8.2.1. Assessment of Causality for Study Drugs and Procedures

The investigator or qualified subinvestigator is responsible for assessing the relationship to IMP therapy using clinical judgment and the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the investigational medicinal product. For SAEs, an alternative causality must be provided (e.g., pre-existing condition, underlying disease, intercurrent illness, or concomitant medication).
- **Yes**: There is reasonable possibility that the event may have been caused by the investigational medicinal product.

It should be emphasized that ineffective treatment should not be considered as causally related in the context of AE reporting.

The relationship to study procedures (e.g., invasive procedures such as venipuncture or biopsy) should be assessed using the following considerations:

- No: Evidence exists that the AE has an etiology other than the study procedure.
- Yes: The adverse event occurred as a result of protocol procedures (eg., venipuncture)

## 8.2.2. Assessment of Severity

The severity grading of AEs will be assessed as Grade 1, 2, 3, or 4 using the GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities (Appendix 3). For AEs associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.

# 8.3. Investigator Requirements and Instructions for Reporting Adverse Events and Serious Adverse Events

All SAEs, regardless of causal relationship, that occur after the subject first consents to participate in the study (ie, signing the informed consent) and throughout the duration of the study, including the protocol-required 24-week post treatment follow-up period, must be reported to the CRF/eCRF database and Gilead Drug Safety and Public Health (DSPH) as instructed. This also includes any SAEs resulting from protocol-mandated procedures performed from screening onwards.

All AEs, regardless of causal relationship, that occur from initiation of study medication until 4 weeks after last administration of study IMP must be reported to the CRF/eCRF database as instructed.

All AEs should be followed up until resolution or until the adverse event is stable, if possible. Gilead Sciences may request that certain AEs be followed beyond the post-treatment follow up period.

Investigators are not obligated to actively seek SAEs after the 24 week post-treatment follow-up period. However, if the investigator learns of any SAEs that occur after this time and the event is deemed relevant to the use of IMP, he/she should promptly document and report the event directly to Gilead DSPH. Gilead DSPH contact information is as follows: Email: Safety\_FC@gilead.com or Fax: +1 (650) 522-5477. All AEs and SAEs will be recorded in the CRF/eCRF database within the timelines outlined in the CRF/eCRF completion guideline.

#### Serious Adverse Event Paper Reporting Process

• All SAEs will be recorded on the serious adverse event report form and submitted by emailing or faxing the report form within 24 hours of the investigator's knowledge of the event to the attention of the designated CRO Pharmacovigilance Representative.

#### Electronic Serious Adverse Event (eSAE) Reporting Process

- All AEs and SAEs will be recorded in the CRF/eCRF database within the timelines outlined in the CRF/eCRF completion guideline.
- Site personnel record all SAE data in the eCRF database and from there transmit the SAE information to Gilead DSPH within 24 hours of the investigator's knowledge of the event. Detailed instructions can be found in the eCRF completion guidelines.
- If for any reason it is not possible to record the SAE information electronically, ie, the eCRF database is not functioning, record the SAE on the paper serious adverse event reporting form and submit within 24 hours as described above.
- As soon as it is possible to do so, any SAE reported via paper must be transcribed into the eCRF Database according to instructions in the eCRF completion guidelines.
- If an SAE has been reported via a paper form because the eCRF database has been locked, no further action is necessary.

Contact information is as follows:

Gilead Sciences, Fax: +1 650 522-5477

Drug Safety and E-mail: Safety FC@gilead.com

Public Health:

CRO Fax: TBD

Pharmacovigilance E-mail:

Representative:

Gilead Sciences, Name: Luisa Stamm, MD, PhD

Medical Monitor: Phone: PPD

Mobile: PPD Fax: PPD E-mail: PPD

- For fatal or life-threatening events, copies of hospital case reports, autopsy reports, and
  other documents are also to be submitted by e-mail or fax when requested and applicable.
  Transmission of such documents should occur without personal subject identification,
  maintaining the traceability of a document to the subject identifiers.
- Additional information may be requested to ensure the timely completion of accurate safety reports.

Any medications necessary for treatment of the SAE must be recorded onto the concomitant medication section of the subject's CRF/eCRF and the event description section of the SAE report form.

#### 8.4. Gilead Reporting Requirements

Depending on relevant local legislation or regulations, including the applicable US FDA Code of Federal Regulations, the EU Clinical Trials Directive (2001/20/EC) and relevant updates, and other country-specific legislation or regulations, Gilead may be required to expedite to worldwide regulatory agencies reports of SAEs, serious adverse drug reactions (SADRs), or suspected unexpected serious adverse reactions (SUSARs). In accordance with the EU Clinical Trials Directive (2001/20/EC), Gilead or a specified designee will notify worldwide regulatory agencies and the relevant IEC in concerned Member States of applicable SUSARs as outlined in current regulations.

Assessment of expectedness for SAEs will be determined by Gilead using reference safety information specified in the investigator's brochure or relevant local label as applicable.

All investigators will receive a safety letter notifying them of relevant SUSAR reports. The investigator should notify the IRB or IEC of SUSAR reports as soon as is practical, where this is required by local regulatory agencies, and in accordance with the local institutional policy.

#### 8.5. Special Situations Reports

### 8.5.1. Definitions of Special Situations

Special situation reports include all reports of medication error, abuse, misuse, overdose, and pregnancy reports regardless of an associated AE. Also includes reports of adverse reactions in infants following exposure from breastfeeding, and reports of adverse reactions associated with product complaints and reports arising from occupational exposure.

A pregnancy report is used to report any pregnancy following maternal or paternal exposure to the medicinal product.

Medication error is any unintentional error in the prescribing, dispensing, or administration of a medicinal product while in the control of the health care provider, subject, or consumer.

Abuse is defined as persistent or sporadic intentional excessive use of a medicinal product by a subject.

Misuse is defined as any intentional and inappropriate use of a medicinal product that is not in accordance with the protocol instructions or the local prescribing information.

An overdose is defined as an accidental or intentional administration of a quantity of a medicinal product given per administration or cumulatively which is above the maximum recommended dose as per protocol or in the product labelling (as it applies to the daily dose of the subject in question). In cases of a discrepancy in drug accountability, overdose will be established only when it is clear that the subject has taken the excess dose(s). Overdose cannot be established when the subject cannot account for the discrepancy except in cases in which the investigator has reason to suspect that the subject has taken the additional dose(s).

Product complaint is defined as complaints arising from potential deviations in the manufacture, packaging or distribution of the medicinal product.

#### 8.5.2. Instructions for Reporting Special Situations

# 8.5.2.1. Instructions for Reporting Pregnancies

The investigator should report all pregnancies that are identified after the subject first consents to participate in the study (ie, signs the informed consent) and throughout the study, including the post-treatment follow-up period, to the CRO Pharmacovigilance Representative using the pregnancy report form within 24 hours of becoming aware of the pregnancy.

The pregnancy itself is not considered an AE nor is an induced elective abortion to terminate a pregnancy without medical reasons.

Any premature termination of pregnancy (eg, a spontaneous abortion, an induced therapeutic abortion due to complications or other medical reasons) must be reported within 24 hours as an SAE. The underlying medical reason for this procedure should be recorded as the AE term.

A spontaneous abortion is always considered to be an SAE and will be reported as described in Sections 8.1.1 and 8.3. Furthermore, any SAE occurring as an adverse pregnancy outcome post study must be reported directly to Gilead DSPH.

The subject should receive appropriate monitoring and care until the conclusion of the pregnancy. The outcome should be reported to CRO Pharmacovigilance Representative using the pregnancy outcome report form. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH. Gilead DSPH contact information is as follows: Email: Safety FC@gilead.com or Fax: +1 (650) 522-5477.

Pregnancies of female partners of male study subjects exposed to Gilead or other study drugs must also be reported and relevant information should be submitted to the CRO Pharmacovigilance Representative using the pregnancy report form and pregnancy outcome report forms within 24 hours. Monitoring of the partner pregnancy should continue until the conclusion of the pregnancy. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH, fax number +1 (650) 522-5477 or email Safety\_FC@gilead.com.

Clinical staff should also report any pregnancies to the Ribavirin Pregnancy Registry at 1-800-593-2214 (see also http://www.ribavirinpregnancyregistry.com).

Refer to Appendix 5 for Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements.

#### 8.5.2.2. Reporting Other Special Situations

All other special situation reports must be reported on the special situations report form and forwarded to the CRO Pharmacovigilance Representative within 24 hours of the investigator

becoming aware of the situation. These reports must consist of situations that involve study IMP, but do not apply to concomitant medications. Except for situations that result in AEs, special situations involving concomitant medications will not be reported. Any inappropriate use of contraindicated medications should not be reported as "misuse," but may be more appropriately documented as a protocol deviation.

Refer to Section 8.3 and the CRF/eCRF completion guidelines for full instructions on the mechanism of special situations reporting.

All clinical sequelae in relation to these special situation reports will be reported as AEs or SAEs at the same time using the AE eCRF and/or the SAE report form. Details of the symptoms and signs, clinical management and outcome will be reported, when available.

## 9. STATISTICAL CONSIDERATIONS

# 9.1. Analysis Objectives and Endpoints

#### 9.1.1. Analysis Objectives

The primary objective of Part A of this study is:

 To evaluate the steady state pharmacokinetics (PK) and confirm the dose of SOF in HCV-infected pediatric subjects

The secondary objective of Part A of this study is:

 To evaluate the safety and tolerability of 7 days of dosing of SOF in HCV-infected pediatric subjects

The primary objectives of Part B of this study are:

- To evaluate the safety and tolerability of SOF + RBV for 12 or 24 weeks in HCV-infected pediatric subjects with genotype 2 or 3, respectively
- To determine the antiviral efficacy of SOF+RBV treatment in genotype 2 and genotype 3 HCV-infected subjects separately, as assessed by the proportion of subjects with SVR 12 weeks after completion of treatment (SVR12)

The secondary objectives of Part B of this study are:

- To determine the antiviral efficacy of SOF+RBV treatment in genotype 2 and genotype 3 HCV-infected subjects separately, as assessed by the proportion of subjects with SVR 4 and 24 weeks after completion of treatment (SVR4 and SVR24)
- To evaluate the kinetics of circulating HCV RNA during treatment and after completion of treatment
- To evaluate the emergence of viral resistance to SOF during treatment and after completion of treatment

The exploratory objective of this study is:



#### 9.1.2. Primary Endpoint

In Part A, AUC<sub>tau</sub> of GS-331007 is considered as the primary PK parameter for determining the appropriate SOF dose.

For Part B, the primary efficacy endpoint is SVR12. Safety endpoint is any AE leading to permanent discontinuation of study drug(s).

#### 9.1.3. Secondary Endpoints

In Part A, the secondary PK endpoints include  $AUC_{tau}$ ,  $C_{max}$ ,  $AUC_{last}$ ,  $T_{max}$ ,  $C_{last}$ ,  $T_{last}$ ,  $C_{tau}$  and  $t_{1/2}$  for GS-331007 and SOF as appropriate. AEs leading to permanent discontinuation of study drug(s) will be evaluated as a secondary safety endpoint.

For Part B, secondary efficacy endpoints include SVR4, SVR24, end-of-treatment response, breakthrough and relapse. Additional efficacy evaluations may include HCV RNA change from Day 1; ALT normalization; viral kinetic parameters; and changes in patient reported outcomes based on the Quality of Life survey to assess the effect of treatment on quality of life.

#### 9.2. Analysis Conventions

All individual subject data will be listed as measured. All statistical summaries and analyses will be performed using SAS® software (SAS Institute, Cary, North Carolina, USA).

## 9.2.1. Analysis Sets

#### 9.2.1.1. Pharmacokinetics (PK) Analysis Sets

#### **Intensive PK Analysis Set**

The intensive PK analysis set will include all part A subjects who received at least one dose of study drug and for whom at least one non-missing PK concentration data, during the intensive sampling period, reported by PK lab. The PK analysis set will be used for detailed pharmacokinetic analysis of SOF, and metabolites.

# **Sparce PK Analysis Set**

The PK analysis set will include all enrolled subjects who received at least one dose of study drug and for whom at least one observed concentration data of SOF or GS-331007 are available. The PK analysis set will be used for analysis of general PK and single sample plasma concentrations.

#### 9.2.1.2. Safety Analysis Set

The primary analysis set for safety analyses will include subjects who were enrolled and have received at least one dose of study drug.

Treatment-emergent data will be analyzed and defined as data collected from the first dose of study drug through the date of last dose of study drug plus 30 days.

#### 9.2.1.3. Efficacy Analysis Set

The analysis set for antiviral activity analyses will be the Full Analysis Set (FAS) which includes HCV infected subjects who were enrolled and have received at least one dose of study drug.

#### 9.2.2. Data Handling Conventions

Natural logarithm transformation for key PK parameters, such as C<sub>max</sub> and AUC<sub>tau</sub>, will be applied for pharmacokinetic analysis.

The PK concentration values below the limit of quantitation (BLQ) will be treated as zero for the determination of summary and order statistics. Individual values that are BLQ will be presented as "BLQ" in the concentration data listing and will be excluded in any calculation of geometric means or ratios. For the presentation of summary and order statistics, if at least 1 subject has a concentration value BLQ for the time point, then the minimum value will be displayed as "BLQ". If more than 50% of the subjects have a concentration data value BLQ for the time point, then the minimum and median values will be displayed as "BLQ". If all subjects have concentration data values BLQ for the time point, then all order statistics (minimum, first quartile [Q1], median, third quartile [Q3], maximum) will be displayed as "BLQ".

Missing data can have an impact upon the interpretation of the trial data. Other than the endpoints discussed below, in general, values for missing data will not be imputed.

For the analysis of post-baseline categorical efficacy endpoints, if a data point is missing and is preceded and followed in time by values that are deem successes, then the missing data point will be termed a success; otherwise the data point will be termed a failure.

Any subject with missing data due to premature discontinuation of the study medication will be considered a failure at the time points subsequent to the date of discontinuation. If no HCV RNA values are obtained after the last dose of study medication, the subject will be considered a treatment failure for the SVR endpoints.

Where appropriate, safety data for subjects that did not complete the study will be included in summary statistics. For example,

- If a subject received study medication, the subject will be included in a summary of adverse events according to the treatment received; otherwise, if the subject is not dosed then they will be excluded from the summary.
- If safety laboratory results for a subject are missing for any reason at a time point, the subject will be excluded from the calculation of summary statistics for that time point. If the subject is missing a pre-dose value, then the subject will be excluded from the calculation of summary statistics for the pre-dose value and the change from pre-dose values.

Values for missing safety laboratory data will not be imputed; however, a missing baseline result will be replaced with a screening result, if available. If no pre-treatment laboratory value is available, the baseline value will be assumed to be normal (i.e., no grade [Grade 0]) for the summary of graded laboratory abnormalities.

Values for missing vital signs data will not be imputed; however, a missing baseline result will be replaced with a screening result, if available.

HCV RNA values below the LLOQ for the assay will be set to the lower limit minus 1 for calculation of summary statistics for the actual HCV RNA values and the change from baseline values by study visit. The reported values will be provided in the HCV RNA listing.

For selected analyses of early time point data, HCV RNA data (IU/mL) may be transformed to the logarithmic (base 10) scale (log<sub>10</sub> IU/mL).

#### 9.2.3. Interim Analysis

No formal interim analyses are planned for this study.

#### 9.3. Demographic Data and Baseline Characteristics

Demographic and baseline measurements will be summarized using standard descriptive methods by age group and overall for Part A and Part B respectively.

Demographic data will include sex, self-identified race/ethnicity, and age.

Baseline characteristic data will include body weight, height, body mass index, HCV RNA level (log<sub>10</sub> IU/mL), HCV genotype, prior treatment experience, and additional endpoints as necessary.

#### 9.4. Pharmacokinetic Analysis

PK analysis will be performed for Part A using the intensive PK analysis set. The concentration data of SOF and metabolites (GS-566500 and GS-331007) over sampling time will be listed and summarized by nominal time and cohort. Pharmacokinetic parameters (e.g., AUC<sub>tau</sub>, AUC<sub>last</sub>, C<sub>max</sub>, T<sub>max</sub>, C<sub>last</sub>, T<sub>last</sub>, C<sub>tau</sub>,  $\lambda z$ , CL/F, Vz/F and  $t^{1}/2$ ) will be listed and summarized for SOF and metabolites (as applicable) using descriptive statistics (e.g., sample size, arithmetic mean, geometric mean and its 95% confidence interval, coefficient of variation %, standard deviation, median, Q1, Q3, minimum, and maximum) by cohort and overall. Plasma concentrations over time will be plotted in semilogarithmic and linear formats as mean  $\pm$  standard deviation, and median (Q1, Q3).

To evaluate the exposures of GS-331007 achieved in pediatric subjects of this study are similar to the exposures observed in historical control subjects, GS-331007 exposure data from this study will be compared to the integrated historical control data by carrying out an analysis of variance (ANOVA) for log-transformed AUC<sub>tau</sub> of GS-331007 as the primary endpoint while C<sub>max</sub> of GS-331007 will be evaluated as secondary endpoints. The 90% confidence intervals will be constructed for the ratio of geometric means of each PK parameters. The equivalence boundary is set as 50% to 200%. Individual patient management will be performed by maintaining exposures comparable to adults. AUCtau less than the 2.5<sup>th</sup> percentile of adult values may require dose adjustment as appropriate.

The effect of age and SOF dose on PK (SOF and GS-331007) will be assessed.

#### 9.5. Efficacy Analysis

Efficacy will be evaluated using scheduled assessments of HCV RNA performed using COBAS® TaqMan® HCV Test, v2.0 for use with the High Pure System.

Efficacy analysis will be performed by age group and genotype for Part B.

All continuous endpoints will be summarized using an 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum). All categorical endpoints will be summarized by number and percentage of subjects who meet the endpoint definition.

#### 9.5.1. Primary Analysis

The primary efficacy endpoint is SVR12 (HCV RNA < LLOQ 12 weeks after completion of treatment) in the FAS population. The primary analysis will be performed after all enrolled subjects have been followed through 12 weeks post-treatment or discontinued from study.

#### 9.5.2. Secondary Analysis

The proportion of subjects with HCV RNA below LLOQ over time (including SVR endpoints) will be presented by age group and genotype in Part B in tabular and graphical form.

Descriptive summaries and listings will be provided for additional efficacy evaluations including serum HCV RNA actual values and change from baseline, proportion of subjects with virologic failures, and other endpoints of interest including ALT normalization.



#### 9.5.3. Subgroup Analysis

Subgroup analysis on SVR24 and SVR12 will be performed by treatment experience (treatment-naive vs. experienced), and by treatment experience and genotype.

Details on efficacy analyses will be described in the statistical analysis plan.

#### 9.6. Safety Analysis

Safety analysis will be performed for Part A and Part B respectively.

Safety will be evaluated by assessment of clinical laboratory tests, physical examinations, vital signs measurements, and by the documentation of AEs.

All safety data collected while on or after the first dose of study drug administration up to 30 days after the last dose of study drug will be summarized by cohort according to the study drug received.

Safety endpoints will be analyzed by the number and percent of subjects with events or abnormalities for categorical values or 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data.

#### 9.6.1. Extent of Exposure

A subject's extent of exposure to study drug will be generated from the study drug administration page of the CRF. Exposure data will be summarized.

#### 9.6.2. Adverse Events

Clinical and laboratory AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC), High-Level Group Term (HLGT), High-Level Term (HLT), Preferred Term (PT), and Lower-Level Term (LLT) will be attached to the clinical database.

Events will be summarized on the basis of the date of onset for the event. A treatment-emergent adverse event will be defined as any new or worsening adverse event that begins on or after the date of first dose of study drug up to the date of last dose of study drug plus 30 days.

Summaries (number and percentage of subjects) of treatment-emergent adverse events (by SOC and preferred term) will be provided by cohort:

- All AEs,
- All study drug-related AEs,
- Combined Grade 2, 3 and 4 AEs,
- Combined Grade 3 and 4 AEs,
- Combined Grade 2, 3 and 4 study drug-related AEs,
- Combined Grade 3 and 4 study drug-related AEs,
- All AEs that caused permanent discontinuation from study drug,
- All AEs that caused change in dose or temporary interruption of study drug,
- All SAEs (including death), and
- All study drug-related SAEs

All AEs collected during the course of the study will be presented in data listings.

#### 9.6.3. Laboratory Evaluations

Selected laboratory data will be summarized using only observed data. Absolute values and changes from baseline at all scheduled visits will be summarized by age group and overall.

Graded laboratory abnormalities will be defined using the grading scheme in Grading of Laboratory Abnormalities provided in Appendix 3.

Incidence of treatment-emergent laboratory abnormalities, defined as values that increase by at least one toxicity grade from baseline at any time post baseline up to and including the date of last dose of study drug plus 30 days, will be summarized by age group and overall. If baseline data are missing, then any graded abnormality (i.e., at least a Grade 1) will be considered treatment emergent.

All laboratory abnormalities will be included in the listings of laboratory data.

#### 9.6.4. Other Safety Evaluations

# 9.6.4.1. Tanner Pubertal Stage Assessment

Tanner Stages (Appendix 4) will be summarized by baseline Tanner Stage using frequency and percentage. Age of first menses will be summarized descriptively.

# 9.7. Data Monitoring Committee

An external multidisciplinary data monitoring committee (DMC) will review the progress of the study and perform interim reviews of safety and PK data and provide recommendation to Gilead about whether the nature, frequency, and severity of adverse effects associated with study treatment warrant the early termination of the study in the best interests of the participants, whether the study should continue as planned, or the study should continue with modifications.

The DMC's specific activities will be defined by a mutually agreed charter, which will define the DMC's membership, conduct and meeting schedule.

While the DMC will be asked to advise Gilead regarding future conduct of the study, including possible early study termination, Gilead retains final decision-making authority on all aspects of the study.

# 9.8. Sample Size

With approximately 50 subjects enrolled into each age group of Part B, a two-sided 95.0% confidence interval of the SVR12 rate will extend at most 11.1% in both directions from the observed SVR12 rate, assuming the expected SVR12 rate is 80%.

## 10. RESPONSIBILITIES

## 10.1. Investigator Responsibilities

#### 10.1.1. Good Clinical Practice

The investigator will ensure that this study is conducted in accordance with the principles of the "Declaration of Helsinki" (as amended in Edinburgh, Tokyo, Venice, Hong Kong, and South Africa), International Conference on Harmonisation (ICH) guidelines, or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the study subject. For studies conducted under a United States IND, the investigator will ensure that the basic principles of "Good Clinical Practice," as outlined in 21 CFR 312, subpart D, "Responsibilities of Sponsors and Investigators," 21 CFR, part 50, 1998, and 21 CFR, part 56, 1998, are adhered to.

Since this is a "covered" clinical trial, the investigator will ensure that 21 CFR, Part 54, 1998, is adhered to; a "covered" clinical trial is any "study of a drug or device in humans submitted in a marketing application or reclassification petition subject to this part that the applicant or FDA relies on to establish that the product is effective (including studies that show equivalence to an effective product) or that make a significant contribution to the demonstration of safety." This requires that investigators and all subinvestigators must provide documentation of their financial interest or arrangements with Gilead Sciences, or proprietary interests in the drug being studied. This documentation must be provided before participation of the investigator and any subinvestigator. The investigator and subinvestigator agree to notify Gilead Sciences of any change to reportable interests during the study and for one year following completion of the study. Study completion is defined as the date that the last subject has completed the protocol defined activities.

This study is also subject to and will be conducted in accordance with 21 CFR, part 320, 1993, "Retention of Bioavailability and Bioequivalence Testing Samples."

# 10.1.2. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) Approval

This protocol and any accompanying material to be provided to the subject (such as advertisements, subject information sheets, or descriptions of the study used to obtain informed consent/assent) will be submitted by the investigator to an IRB (for studies conducted in the United States) or IEC (for studies conducted outside of the United States). Approval from the IRB or IEC must be obtained **before** starting the study and should be documented in a letter to the investigator specifying the protocol number, protocol version, protocol date, documents reviewed, and date on which the committee met and granted the approval.

Any modifications made to the protocol after receipt of IRB or IEC approval must also be submitted to the IRB or IEC for approval before implementation.

#### 10.1.3. Informed Consent/Assent

The investigator is responsible for obtaining written informed consent from the parent/legal guardian of the subject participating in this study after adequate explanation to the parent/legal guardian and subject of the aims, methods, objectives, and potential hazards of the study and before undertaking any study-related procedures. Written assent should be obtained from the subject as required by IRB/IEC/local requirements for this age population. The investigator must utilize an IRB- or IEC-approved consent/assent form for documenting written informed consent/assent. Each informed consent/assent will be appropriately signed and dated by the subject or the subject's parent/legally authorized representative and the person obtaining consent/assent.

#### 10.1.4. Confidentiality

The investigator must assure that subjects' anonymity will be strictly maintained and that their identities are protected from unauthorized parties. Only subject initials, date of birth, and an identification code (i.e., not names) should be recorded on any form or biological sample submitted to the Sponsor, IRB or IEC, or laboratory. The investigator must keep a screening log showing codes, names, and addresses for all subjects screened and for all subjects enrolled in the trial.

The investigator agrees that all information received from Gilead Sciences, including but not limited to the Investigator Brochure, this protocol, CRFs, the investigational new drug, and any other study information, remain the sole and exclusive property of Gilead Sciences during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from Gilead Sciences. The investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

#### 10.1.5. Study Files and Retention of Records

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into at least the following two categories: (1) investigator's study file, and (2) subject clinical source documents.

The investigator's study file will contain the protocol/amendments, CRF and query forms, IRB or IEC and governmental approval with correspondence, informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

The required source data are listed in the Source Data verification Plan, and should include sequential notes containing at least the following information for each subject:

- Subject identification (name, date of birth, gender);
- Documentation that subject meets eligibility criteria, i.e., history, physical examination, and confirmation of diagnosis (to support inclusion and exclusion criteria);
- Participation in trial (including trial number);
- Trial discussed and date of informed consent;
- Dates of all visits;
- Documentation that protocol specific procedures were performed;
- Results of efficacy parameters, as required by the protocol;
- Start and end date (including dose regimen) of trial medication (preferably drug dispensing and return should be documented as well);
- Record of all AEs and other safety parameters (start and end date, and preferably including causality and intensity);
- Concomitant medication (including start and end date, dose if relevant; dose changes should be motivated);
- Date of trial completion and reason for early discontinuation, if applicable.

All clinical study documents must be retained by the investigator until at least 2 years after the last approval of a marketing application in an ICH region (i.e., United States, Europe, or Japan) and until there are no pending or contemplated marketing applications in an ICH region; or, if no application is filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and regulatory authorities have been notified. Investigators may be required to retain documents longer if required by applicable regulatory requirements, by local regulations, or by an agreement with Gilead Sciences. The investigator must notify Gilead Sciences before destroying any clinical study records.

Should the investigator wish to assign the study records to another party or move them to another location, Gilead Sciences must be notified in advance.

If the investigator cannot guarantee this archiving requirement at the study site for any or all of the documents, special arrangements must be made between the investigator and Gilead Sciences to store these in sealed containers outside of the site so that they can be returned sealed to the investigator in case of a regulatory audit. When source documents are required for the continued care of the subject, appropriate copies should be made for storage outside of the site.

Biological samples at the conclusion of this study may be retained in storage by the Sponsor for a period up to 10 years for purposes of this study.

### 10.1.6. Case Report Forms

For each subject enrolled, a CRF (or eCRF) must be completed and signed by the principal investigator or subinvestigator (as appropriate) within a reasonable time period after data collection. This also applies to records for those subjects who fail to complete the study (even during a prerandomization screening period if a CRF was initiated). If a subject withdraws from the study, the reason must be noted on the CRF. If a subject is withdrawn from the study because of a treatment-limiting adverse event, thorough efforts should be made to clearly document the outcome.

# 10.1.7. Drug Accountability

The investigator or designee (i.e., pharmacist) is responsible for ensuring adequate accountability of all used and unused investigational medicinal product, and comparators. This includes acknowledgment of receipt of each shipment of study product (quantity and condition), subject dispensing records, and returned or destroyed study product. Dispensing records will document quantities received from Gilead Sciences and quantities dispensed to subjects, including lot number, date dispensed, subject identifier number, subject initials, and the initials of the person dispensing the medication.

At study initiation, the monitor will evaluate the site's standard operating procedure for investigational medicinal product disposal/destruction in order to ensure that it complies with Gilead Sciences requirements. Drug may be returned or destroyed on an ongoing basis during the study if appropriate. At the end of the study, following final drug inventory reconciliation by the monitor, the study site will dispose of and/or destroy all unused investigational medicinal product supplies, including empty containers, according to these procedures. If the site cannot meet Gilead Sciences' requirements for disposal, arrangements will be made between the site and Gilead Sciences or its representative for destruction or return of unused investigational medicinal product supplies.

All drug supplies and associated documentation will be periodically reviewed and verified by the study monitor over the course of the study.

#### 10.1.8. Inspections

The investigator should understand that source documents for this trial should be made available to appropriately qualified personnel from Gilead Sciences or its representatives, to IRBs or IECs, or to regulatory authority or health authority inspectors.

# 10.1.9. Protocol Compliance

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol.

#### 10.2. Sponsor Responsibilities

#### 10.2.1. Protocol Modifications

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by Gilead Sciences. All protocol modifications must be submitted to the IRB or IEC in accordance with local requirements. Approval must be obtained before changes can be implemented.

#### 10.2.2. Study Report and Publications

A clinical study report will be prepared and provided to the regulatory agency(ies). Gilead Sciences will ensure that the report meets the standards set out in the ICH Guideline for Structure and Content of Clinical Study Reports (ICH E3). Note that an abbreviated report may be prepared in certain cases.

After conclusion of the study and without prior written approval from Gilead Sciences, investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media *only after the following conditions have been met:* 

- the results of the study in their entirety have been publicly disclosed by or with the consent of Gilead Sciences in an abstract, manuscript, or presentation form; or
- the study has been completed at all study sites for at least 2 years.

No such communication, presentation, or publication will include Gilead Sciences' confidential information (see Section 10.1.4).

The investigator will submit any proposed publication or presentation along with the respective scientific journal or presentation forum at least 30 days before submission of the publication or presentation. The investigator will comply with Gilead Sciences' request to delete references to its confidential information (other than the study results) in any paper or presentation and agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.

# 10.3. Joint Investigator/Sponsor Responsibilities

#### **10.3.1.** Access to Information for Monitoring

In accordance with ICH Good Clinical Practice (ICH GCP) guidelines, the study monitor must have direct access to the investigator's source documentation in order to verify the data recorded in the CRFs for consistency.

The monitor is responsible for routine review of the CRFs at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The monitor should have access to any subject records needed to verify the entries on the CRFs. The investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits are resolved.

#### **10.3.2.** Access to Information for Auditing or Inspections

Representatives of regulatory authorities or of Gilead Sciences may conduct inspections or audits of the clinical study. If the investigator is notified of an inspection by a regulatory authority the investigator agrees to notify the Gilead Sciences medical monitor immediately. The investigator agrees to provide to representatives of a regulatory agency or Gilead Sciences access to records, facilities, and personnel for the effective conduct of any inspection or audit.

## 10.3.3. Study Discontinuation

Both the sponsor and the investigator reserve the right to terminate the study at any time. Should this be necessary, both parties will arrange discontinuation procedures and notify the appropriate regulatory authority(ies), IRBs, and IECs. In terminating the study, Gilead Sciences and the investigator will assure that adequate consideration is given to the protection of the subjects' interests.

## 11. REFERENCES

- Poynard T, Marcellin P, Lee SS, Niederau C, Minuk GS, Ideo G, et al. Randomised trial of interferon alpha2b plus ribavirin for 48 weeks or for 24 weeks versus interferon alpha2b plus placebo for 48 weeks for treatment of chronic infection with hepatitis C virus. International Hepatitis Interventional Therapy Group (IHIT). Lancet 1998;352 (9138):1426-32.
- McHutchison JG, Gordon SC, Schiff ER, Shiffman ML, Lee WM, Rustgi VK, et al. Interferon alfa-2b alone or in combination with ribavirin as initial treatment for chronic hepatitis C. Hepatitis Interventional Therapy Group. N Engl J Med 1998;339 (21):1485-92.
- 15572 COPEGUS® (ribavirin, USP) TABLETS. US Prescribing Information. Roche Laboratories Inc., Nutley, NJ. Revised: January 2010.
- Copegus 200mg and 400mg Film-coated Tablets. Summary of Product Characteristics. Roche Products Limited, Welwyn Garden City, United Kingdom. Revised: March 2010.
- Esteban JI, Sauleda S, Quer J. The changing epidemiology of hepatitis C virus infection in Europe. J Hepatol 2008;48 (1):148-62.
- Hu J, Doucette K, Hartling L, Tjosvold L, Robinson J. Treatment of hepatitis C in children: a systematic review. PLoS ONE 2010;5 (7):e11542.
- Mohan N, Gonzalez-Peralta RP, Fujisawa T, Chang MH, Heller S, Jara P, et al. Chronic hepatitis C virus infection in children. J Pediatr Gastroenterol Nutr 2010;50 (2):123-31.
- 20273 Bortolotti F, Verucchi G, Camma C, Cabibbo G, Zancan L, Indolfi G, et al. Long-term course of chronic hepatitis C in children: from viral clearance to end-stage liver disease. Gastroenterology 2008;134 (7):1900-7.
- 20282 Serranti D, Buonsenso D, Ceccarelli M, Gargiullo L, Ranno O, Valentini P. Pediatric hepatitis C infection: to treat or not to treat...what's the best for the child? European review for medical and pharmacological sciences 2011;15 (9):1057-67.
- Wirth S. Current treatment options and response rates in children with chronic hepatitis C. World J Gastroenterol 2012;18 (2):99-104.
- Wirth S, Ribes-Koninckx C, Calzado MA, Bortolotti F, Zancan L, Jara P, et al. High sustained virologic response rates in children with chronic hepatitis C receiving peginterferon alfa-2b plus ribavirin. J Hepatol 2010;52 (4):501-7.
- Zhu HJ, Appel DI, Jiang Y, Markowitz JS. Age- and sex-related expression and activity of carboxylesterase 1 and 2 in mouse and human liver. Drug Metab Dispos 2009;37 (9):1819-25.
- Gane EJ, Stedman CA, Hyland RH, Ding X, Svarovskaia E, Symonds WT, et al. Nucleotide polymerase inhibitor sofosbuvir plus ribavirin for hepatitis C. N Engl J Med 2013;368 (1):34-44.
- Jacobson IM, Gordon SC, Kowdley KV, Yoshida EM, Rodriguez-Torres M, Sulkowski MS, et al. Sofosbuvir for hepatitis C genotype 2 or 3 in patients without treatment options. N Engl J Med 2013;368 (20):1867-77.
- 24715 Lawitz E, Mangia A, Wyles D, Rodriguez-Torres M, Hassanein T, Gordon SC, et al. Sofosbuvir for previously untreated chronic hepatitis C infection. N Engl J Med 2013;368 (20):1878-87.
- SOVALDI™ (sofosbuvir) tablets, for oral use. US Prescribing Information. Gilead Sciences, Inc. Foster City, CA. December 2013.

# 12. APPENDICES

| Appendix 1. | Investigator Signature Page |
|-------------|--------------------------------------------------------------|
| Appendix 2. | Study Procedures Table |
| Appendix 3. | GSI Grading Scale for Severity of Adverse Events and |
| | Laboratory Abnormalities |
| Appendix 4. | Tanner Stages |
| Appendix 5. | Pregnancy Precautions, Definition for Female of Childbearing |
| | Potential, and Contraceptive Requirements |

Date

#### Appendix 1. **Investigator Signature Page**

# GILEAD SCIENCES, INC. 333 LAKESIDE DRIVE **FOSTER CITY, CA 94404**

### STUDY ACKNOWLEDGEMENT

A Phase 2 Open-Label Multicenter Multi-cohort Single-Arm Study to Investigate the

| Safety and Efficacy of Sofosbuvir + Ribavirin in Adolescents and Children with Genotype 2 or 3 Chronic HCV Infection |
|---|
| GS-US-334-1112, Original, 20 December 2013 |
| This protocol has been approved by Gilead Sciences, Inc. The following signature documents this approval. |
| PPD |
| Luisa Stamm |
| Luisa Stamm, MD, Ph.D (Printed) Medical Monitor Sig |
| 12.23.13 |
| Date |
| INVESTIGATOR STATEMENT |
| I have read the protocol, including all appendices, and I agree that it contains all necessary details for me and my staff to conduct this study as described. I will conduct this study as outlined herein and will make a reasonable effort to complete the study within the time designated. |
| I will provide all study personnel under my supervision copies of the protocol and access to all information provided by Gilead Sciences, Inc. I will discuss this material with them to ensure that they are fully informed about the drugs and the study. |
| Principal Investigator Name (Printed) Signature |

Site Number

**Appendix 2. Study Procedures Table** 

# Appendix Table 1. Part A: Screening and On-Treatment Study Visits

| | | On-treatment | | |
|---|---|---|---|---|
| | Screening<br>(-28 days) | Day 1 <sup>b</sup> | Day 3 | <b>Day 7</b> (+ 3 days) |
| Clinical Assessments | · | | | |
| Informed Consent / Assent | X | | | |
| Determine Eligibility | X | X | | |
| Medical History | X | | | |
| Complete Physical Examination | X | X | | |
| Symptom-directed Physical Examination | | | X | X |
| Tanner Pubertal Stage Assessment | X | | | |
| Vital Signs <sup>a</sup> | X | X | X | X |
| AEs and Concomitant Medications | X | X | X | X |
| Pregnancy Prevention Counseling <sup>f</sup> | | X | | |
| SOF Swallowability Assessment | | X | | |
| Review of Study<br>Medication Compliance | | | | X |
| Study Drug Dispensing <sup>b</sup> | | X | | |
| Laboratory Assessments | | <u>.</u> | | |
| Hematology, Chemistry | X | X | X | X |
| Coagulation Tests | X | X | | |

| | | | On-treatment | |
|---|---|---|---|---|
| | Screening<br>(-28 days) | Day 1 <sup>b</sup> | Day 3 | Day 7<br>(+ 3 days) |
| HCV RNA | X | X | X | X |
| Viral Sequencing <sup>c</sup> | | X | X | X |
| Serum or Urine Pregnancy Testing <sup>e</sup> | X | X | | X |
| Urinalysis | X | X | | X |
| Urine Drug Screen | X | | | |
| Intensive PK | | | | X <sup>d</sup> |
| HCV Genotyping, IL28B | X | | | |
| HCV antibody, HIV 1/2 antibody, HBs antigen, HAV antibody | X | | | |
| HbA1c | X | | | |
| TSH | X | | | |
| Alpha fetoprotein | X | | | |
| Alpha-1 anti-trypsin | X | | | |

a Vital signs include height, weight, blood pressure, pulse, respiratory rate and temperature

b Day 1 assessments must be performed prior to dosing

c Plasma samples will be collected and stored for potential HCV sequencing and other virology studies

d For Cohorts 1 and 2, plasma samples will be collected for PK analyses following dosing of study drugs on Day 7 at the following time points: 0 (predose), 0.5, 1, 2, 3, 4, 8, and 12 hours post-dose. For Cohort 3, plasma samples for PK analyses will be collected at the following time points: 0 (predose), 2, 4, 8, and 12 hours post-dose.

e Females of childbearing potential only. Serum pregnancy test performed at screening and for confirmation of positive urine pregnancy test.

f Including partner pregnancy prevention for male participants (subjects 12 to < 18 years of age only).

# **Appendix Table 2.** Part B: Screening and On-Treatment Study Visits

| | | | Visit identified by on-treatment study week | | | | | | | week | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Day 1 <sup>c</sup> | 1 | 2 | 4 | 8 | 12 | 16 <sup>g</sup> | 20 <sup>g</sup> | 24 <sup>g</sup> | Early<br>Termination |
| Clinical Assessments | | | | | | | | | | | |
| Informed Consent / Assent | X | | | | | | | | | | |
| Determine Eligibility | X | X | | | | | | | | | |
| Medical History | X | | | | | | | | | | |
| Complete Physical Examination | X | X | | | | | X | | | X | X |
| Symptom-Directed Physical Examination | | | X | X | X | X | | X | X | | |
| Tanner Pubertal Stage Assessment & Rates of growth <sup>h</sup> | | X | | | | | X | | | X | X |
| Vital Signs <sup>a</sup> | X | X | X | X | X | X | X | X | X | X | X |
| AEs and Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy Prevention Counseling <sup>i</sup> | | X | | | | | X | | | X | X |
| SOF Swallowability Assessment | | X | | | | | | | | | |
| Quality of Life Survey <sup>e</sup> | | X | | | | | X | | | X | X |
| Review of Study<br>Medication Compliance | | | | | X | X | X | X | X | X | X |
| Study Drug Dispensing <sup>b</sup> | | X | | | X | X | X | X | X | | |
| Laboratory Assessments | | • | | • | • | • | • | • | • | • | • |
| Hematology, Chemistry Coagulation | X | X | X | X | X | X | X | X | X | X | X |
| HCV RNA | X | X | X | X | X | X | X | X | X | X | X |
| Viral Sequencing d | | X | X | X | X | X | X | X | X | X | X |

| | | Visit identified by on-treatment st | | | | | nt study | week | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Day 1 <sup>c</sup> | 1 | 2 | 4 | 8 | 12 | 16 <sup>g</sup> | 20 <sup>g</sup> | 24 <sup>g</sup> | Early<br>Termination |
| Serum or Urine Pregnancy Testing | X | X | | | X | X | X | X | X | X | X |
| Single PK | | | X | X | X | X | X | X | X | X | X |
| PPD | | | | • | | | • | | | | |
| Urinalysis, Urine Drug Test | X | | | | | | | | | | |
| HCV Genotyping, IL28B | X | | | | | | | | | | |
| HCV antibody, HIV 1/2 antibody, HBs antigen, HAV antibody | X | | | | | | | | | | |
| HbA1c | X | | | | | | | | | | |
| TSH | X | | | | | | X | | | X | X |
| Alpha fetoprotein, Alpha-1 anti-trypsin | X | | | | | | | | | | |

- a Vital signs include height, weight, blood pressure, pulse, respiratory rate and temperature
- b The IWRS will provide direction on the specifics of each subject's study drug dispensing.
- c Day 1 assessments must be performed prior to dosing
- d Plasma samples will be collected and stored for potential HCV sequencing and other virology studies
- e Quality of life survey will be completed by all subjects at Day 1, 12, and 24/ET visits if a site is approved to use the survey. Subject is to review questionnaire with a parent/guardian and write/mark answers directly onto the questionnaire.
- f PPD
- g GT-2 subjects will complete through the Week 12 visit; GT-3 subjects will complete through the Week 24 visit.
- h Performed at Day 1 and End of Treatment
- I Including partner pregnancy prevention for male participants (subjects 12 to < 18 years of age only).

# Appendix Table 3. Part B: Post Treatment Visits Following Primary Study

| | 4 Weeks Post Treatment | 12 Weeks Post Treatment | 24 Weeks Post Treatment |
|---|---|---|---|
| Clinical Assessments | | | |
| Vital Signs, Body weight and Height | X | X | X |
| Symptom-directed Physical Exam | X | X | X |
| AEs | X | $X^d$ | $X^d$ |
| Concomitant Medications | X | | |
| Quality of Life Survey <sup>a</sup> | | X | X |
| Tanner Pubertal Stage Assessment & Rates of Growth | | X | X |
| Pregnancy Prevention Counseling <sup>e</sup> | X | X | X |
| Laboratory Assessments | | | |
| Hematology, Chemistry | X | X | |
| HCV RNA | X | X | X |
| Viral Sequencing <sup>b</sup> | X | X | X |
| Urine Pregnancy Test <sup>c</sup> | X | X | X |

a Quality of life survey will be completed by all subjects at 12-Week and 24-Week Post Treatment visits if a site is approved to use the survey. Subject is to review questionnaire with a parent/guardian and write/mark answers directly onto the questionnaire.

b Plasma samples will be collected and stored for potential HCV sequencing and other virology studies

Female subjects of childbearing potential should be provided with Urine Pregnancy Test Kits, instructed on their use and requested to continue to self-monitor for pregnancy for 6 months after their last dose of RBV. If required by regulations, additional pregnancy tests beyond 6 months may be added. The subject should be contacted every 4 weeks and asked to report results of the urine pregnancy tests. If a positive urine pregnancy test is reported, the subject should return to the clinic for a serum pregnancy test.

d All SAEs, including deaths, regardless of cause or relationship, must be reported after patient signs the informed consent through the end of the study

e Including partner pregnancy prevention for male participants (subjects 12 to < 18 years of age only).

Appendix 3. GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities

Version: 18June2012

| | HEMATOLOGY | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin<br>HIV POSITIVE | 8.5 to 10.0 g/dL | 7.5 to < 8.5 g/dL | 6.5 to < 7.5 g/dL | < 6.5 g/dL |
| Adult and Pediatric ≥ 57 Days | 85 to 100 g/L | 75 to < 85 g/L | 65 to < 75 g/L | < 65 g/L |
| HIV NEGATIVE | 10.0 to 10.9 g/dL | 9.0 to < 10.0 g/dL | 7.0 to < 9.0 g/dL | < 7.0 g/dL |
| Adult and Pediatric ≥ 57 Days | 100 to 109 g/L | 90 to < 100 g/L | 70 to < 90 g/L | < 70 g/L |
| | OR | OR | OR | |
| | Any decrease from Baseline | Any decrease from Baseline | Any decrease from Baseline | |
| | 2.5 to < 3.5 g/dL | 3.5 to < 4.5 g/dL | $\geq 4.5 \text{ g/dL}$ | |
| | 25 to < 35 g/L | 35 to < 45 g/L | ≥ 45 g/L | |
| Infant, 36–56 Days | 8.5 to 9.4 g/dL | 7.0 to < 8.5 g/dL | 6.0 to < 7.0 g/dL | < 6.0 g/dL |
| (HIV <u>POSITIVE</u> OR <u>NEGATIVE</u> ) | 85 to 94 g/L | 70 to < 85 g/L | 60 to < 70 g/L | < 60 g/L |
| Infant, 22–35 Days | 9.5 to 10.5 g/dL | 8.0 to < 9.5 g/dL | 7.0 to < 8.0 g/dL | < 7.0 g/dL |
| (HIV <u>POSITIVE</u> OR <u>NEGATIVE</u> ) | 95 to 105 g/L | 80 to < 95 g/L | 70 to < 80 g/L | < 70 g/L |
| Infant, 1–21 Days | 12.0 to 13.0 g/dL | 10.0 to < 12.0 g/dL | 9.0 to < 10.0 g/dL | < 9.0 g/dL |
| (HIV <u>POSITIVE</u> OR <u>NEGATIVE</u> ) | 120 to 130 g/L | 100 to < 120 g/L | 90 to < 100 g/L | < 90 g/L |

| | HEMATOLOGY | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Absolute Neutrophil Count (ANC) | 1000 to 1300/mm <sup>3</sup> | 750 to < 1000/mm <sup>3</sup> | 500 to < 750/mm <sup>3</sup> | < 500/mm <sup>3</sup> |
| Adult and Pediatric, > 7 Days | 1.00 to 1.30 GI/L | 0.75 to < 1.00 GI/L | 0.50 to < 0.75 GI/L | < 0.50 GI/L |
| Infant, 2 – ≤ 7 Days | 1250 to 1500/mm <sup>3</sup> | 1000 to < 1250/mm <sup>3</sup> | 750 to < 1000/mm <sup>3</sup> | < 750/mm <sup>3</sup> |
| | 1.25 to 1.50 GI/L | 1.00 to < 1.25 GI/L | 0.75 to < 1.00 GI/L | < 0.75 GI/L |
| Infant, 1 Day | 4000 to 5000/mm <sup>3</sup> | $3000 \text{ to} < 4000/\text{mm}^3$ | $1500 \text{ to} < 3000/\text{mm}^3$ | < 1500/mm <sup>3</sup> |
| | 4.00 to 5.00 GI/L | 3.00 to < 4.00 GI/L | 1.50 to < 3.00 GI/L | < 1.50 GI/L |
| Absolute CD4+ Count | | | | |
| HIV NEGATIVE ONLY | | | | |
| Adult and Pediatric > 13 Years | 300 to 400/mm <sup>3</sup> | 200 to < 300/mm <sup>3</sup> | $100 \text{ to} < 200/\text{mm}^3$ | < 100/mm <sup>3</sup> |
| > 13 Tears | 300 to 400/μL | $200 \text{ to} < 300/\mu\text{L}$ | $100 \text{ to} < 200/\mu\text{L}$ | < 100/μL |
| Absolute Lymphocyte Count | | | | |
| HIV NEGATIVE ONLY | | | | |
| Adult and Pediatric | 600 to 650/mm <sup>3</sup> | 500 to < 600/mm <sup>3</sup> | 350 to < 500/mm <sup>3</sup> | < 350/mm <sup>3</sup> |
| > 13 Years | 0.60 to 0.65 GI/L | 0.50 to < 0.60 GI/L | 0.35 to < 0.50 GI/L | < 0.35 GI/L |

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Platelets | 100,000 to < 125,000/mm <sup>3</sup> | 50,000 to < 100,000/mm <sup>3</sup> | 25,000 to < 50,000/mm <sup>3</sup> | < 25,000/mm <sup>3</sup> |
| | 100 to < 125 GI/L | 50 to < 100 GI/L | 25 to < 50 GI/L | < 25 GI/L |
| WBCs | 2000/mm <sup>3</sup> to 2500/mm <sup>3</sup> | 1,500 to < 2,000/mm <sup>3</sup> | 1000 to < 1,500/mm <sup>3</sup> | < 1000/mm <sup>3</sup> |
| | 2.00 GI/L to 2.50 GI/L | 1.50 to < 2.00 GI/L | 1.00 to < 1.50 GI/L | < 1.00 GI/L |
| Hypofibrinogenemia | 100 to 200 mg/dL | 75 to < 100 mg/dL | 50 to < 75 mg/dL | < 50 mg/dL |
| | 1.00 to 2.00 g/L | 0.75 to < 1.00 g/L | 0.50 to < 0.75 g/L | < 0.50 g/L |
| Hyperfibrinogenemia | > ULN to 600 mg/dL | > 600 mg/dL | _ | _ |
| | > ULN to 6.0 g/L | > 6.0 g/L | _ | _ |
| Fibrin Split Product | 20 to 40 μg/mL | > 40 to 50 μg/mL | > 50 to 60 μg/mL | > 60 μg/mL |
| | 20 to 40 mg/L | > 40 to 50 mg/L | > 50 to 60 mg/L | > 60 mg/L |
| Prothrombin Time (PT) | > 1.00 to 1.25 × ULN | > 1.25 to 1.50 × ULN | > 1.50 to 3.00 × ULN | > 3.00 × ULN |
| International Normalized Ratio of prothrombin time (INR) | 1.1 to 1.5 x ULN | >1.5 to 2.0 x ULN | >2.0 to 3.0 x ULN | >3.0 x ULN |
| Activated Partial | | | | |
| Thromboplastin Time (APTT) | > 1.00 to 1.66 × ULN | > 1.66 to 2.33 × ULN | > 2.33 to 3.00 × ULN | > 3.00 × ULN |
| Methemoglobin | 5.0 to 10.0% | > 10.0 to 15.0% | > 15.0 to 20.0% | > 20.0% |

| | | CHEMISTRY | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 to <lln l<="" meq="" td=""><td>125 to &lt; 130 mEq/L</td><td>121 to &lt; 125 mEq/L</td><td>&lt; 121 mEq/L</td></lln> | 125 to < 130 mEq/L | 121 to < 125 mEq/L | < 121 mEq/L |
| | 130 to <lln l<="" mmol="" td=""><td>125 to &lt; 130 mmol/L</td><td>121 to &lt; 125 mmol/L</td><td>&lt; 121 mmol/L</td></lln> | 125 to < 130 mmol/L | 121 to < 125 mmol/L | < 121 mmol/L |
| Hypernatremia | 146 to 150 mEq/L | > 150 to 154 mEq/L | > 154 to 159 mEq/L | > 159 mEq/L |
| | 146 to 150 mmol/L | > 150 to 154 mmol/L | > 154 to 159 mmol/L | > 159 mmol/L |
| Hypokalemia | 3.0 to 3.4 mEq/L | 2.5 to < 3.0 mEq/L | 2.0 to < 2.5 mEq/L | < 2.0 mEq/L |
| | 3.0 to 3.4 mmol/L | 2.5 to < 3.0 mmol/L | 2.0 to < 2.5 mmol/L | < 2.0 mmol/L |
| Hyperkalemia | 5.6 to 6.0 mEq/L | > 6.0 to 6.5 mEq/L | > 6.5 to 7.0 mEq/L | > 7.0 mEq/L |
| | 5.6 to 6.0 mmol/L | > 6.0 to 6.5 mmol/L | > 6.5 to 7.0 mmol/L | > 7.0 mmol/L |
| Hypoglycemia | | | | |
| Adult and Pediatric | 55 to 64 mg/dL | 40 to < 55 mg/dL | 30 to < 40 mg/dL | < 30 mg/dL |
| ≥ 1 Month | 3.03 to 3.58 mmol/L | 2.20 to < 3.03 mmol/L | 1.64 to < 2.20 mmol/L | < 1.64 mmol/L |
| Infant, < 1 Month | 50 to 54 mg/dL | 40 to < 50 mg/dL | 30 to < 40 mg/dL | < 30 mg/dL |
| | 2.8 to 3.0 mmol/L | 2.2 to < 2.8 mmol/L | 1.7 to < 2.2 mmol/L | < 1.7 mmol/L |
| Hyperglycemia, Nonfasting | 116 to 160 mg/dL | > 160 to 250 mg/dL | > 250 to 500 mg/dL | > 500 mg/dL |
| | 6.42 to 8.91 mmol/L | > 8.91 to 13.90 mmol/L | > 13.90 to 27.79 mmol/L | > 27.79 mmol/L |
| Hyperglycemia, Fasting | 110 to 125 mg/dL | >125 to 250 mg/dL | >250 to 500 mg/dL | >500 mg/dL |
| | 6.08 to 6.96 mmol/L | >6.96 to 13.90 mmol/L | >13.90 to 27.79 mmol/L | >27.79 mmol/L |

| | CHEMISTRY | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypocalcemia | | | | |
| (corrected for albumin if appropriate*) | 7.8 to 8.4 mg/dL | 7.0 to < 7.8 mg/dL | 6.1 to < 7.0 mg/dL | < 6.1 mg/dL |
| Adult and Pediatric | 1.94 to 2.10 mmol/L | 1.74 to < 1.94 mmol/L | 1.51 to < 1.74 mmol/L | < 1.51 mmol/L |
| ≥7 Days | | | | |
| Infant, < 7 Days | 6.5 to 7.5 mg/dL | 6.0 to < 6.5 mg/dL | 5.5 to < 6.0 mg/dL | < 5.5 mg/dL |
| | 1.61 to 1.88 mmol/L | 1.49 to < 1.61 mmol/L | 1.36 to < 1.49 mmol/L | < 1.36 mmol/L |
| Hypercalcemia (corrected for albumin if appropriate*) | | | | |
| Adult and Pediatric ≥ | >ULN to 11.5 mg/dL | > 11.5 to 12.5 mg/dL | > 12.5 to 13.5 mg/dL | > 13.5 mg/dL |
| 7 Days | >ULN to 2.88 mmol/L | > 2.88 to 3.13 mmol/L | > 3.13 to 3.38 mmol/L | > 3.38 mmol/L |
| Infant, < 7 Days | 11.5 to 12.4 mg/dL | > 12.4 to 12.9 mg/dL | > 12.9 to 13.5 mg/dL | > 13.5 mg/dL |
| | 2.86 to 3.10 mmol/L | > 3.10 to 3.23 mmol/L | > 3.23 to 3.38 mmol/L | > 3.38 mmol/L |
| Hypocalcemia (ionized) | 3.0 mg/dL to < LLN | 2.5 to < 3.0 mg/dL | 2.0 to < 2.5 mg/dL | < 2.0 mg/dL |
| | 0.74 mmol/L to < LLN | 0.62 to < 0.74 mmol/L | 0.49 to < 0.62 mmol/L | < 0.49 mmol/L |
| Hypercalcemia (ionized) | > ULN to 6.0 mg/dL | > 6.0 to 6.5 mg/dL | > 6.5 to 7.0 mg/dL | > 7.0 mg/dL |
| | > ULN to 1.50 mmol/L | > 1.50 to 1.63 mmol/L | > 1.63 to 1.75 mmol/L | > 1.75 mmol/L |
| Hypomagnesemia | 1.40 to <lln dl<="" mg="" td=""><td>1.04 to &lt; 1.40 mg/dL</td><td>0.67 to &lt; 1.04 mg/dL</td><td>&lt; 0.67 mg/dL</td></lln> | 1.04 to < 1.40 mg/dL | 0.67 to < 1.04 mg/dL | < 0.67 mg/dL |
| | 1.2 to <lln l<="" meq="" td=""><td>0.9 to &lt; 1.2 mEq/L</td><td>0.6 to &lt; 0.9 mEq/L</td><td>&lt; 0.6 mEq/L</td></lln> | 0.9 to < 1.2 mEq/L | 0.6 to < 0.9 mEq/L | < 0.6 mEq/L |
| | 0.58 to <lln l<="" mmol="" td=""><td>0.43 to &lt; 0.58 mmol/L</td><td>0.28 to &lt; 0.43 mmol/L</td><td>&lt; 0.28 mmol/L</td></lln> | 0.43 to < 0.58 mmol/L | 0.28 to < 0.43 mmol/L | < 0.28 mmol/L |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypophosphatemia | | | | |
| Adult and Pediatric | 2.0 to < LLN mg/dL | 1.5 to < 2.0 mg/dL | 1.0 to < 1.5 mg/dL | < 1.0 mg/dL |
| > 14 Years | 0.63 to < LLN mmol/L | 0.47 to < 0.63 mmol/L | 0.31 to < 0.47 mmol/L | < 0.31 mmol/L |
| Pediatric 1 Year-14 Years | 3.0 to 3.5 mg/dL | 2.5 to < 3.0 mg/dL | 1.5 to < 2.5 mg/dL | < 1.5 mg/dL |
| | 0.96 to 1.14 mmol/L | 0.80 to < 0.96 mmol/L | 0.47 to < 0.80 mmol/L | < 0.47 mmol/L |
| Pediatric < 1 Year | 3.5 to 4.5 mg/dL | 2.5 to < 3.5 mg/dL | 1.5 to < 2.5 mg/dL | < 1.5 mg/dL |
| | 1.12 to 1.46 mmol/L | 0.80 to < 1.12 mmol/L | 0.47 to < 0.80 mmol/L | < 0.47 mmol/L |
| Hyperbilirubinemia | | | | |
| Adult and Pediatric > 14 Days | > 1.0 to 1.5 × ULN | > 1.5 to 2.5 × ULN | > 2.5 to 5.0 × ULN | > 5.0 × ULN |
| Infant, ≤ 14 Days | NA | 20.0 to 25.0 mg/dL | > 25.0 to 30.0 mg/dL | > 30.0 mg/dL |
| (non-hemolytic) | | 342 to 428 μmol/L | > 428 to 513 μmol/L | > 513 μmol/L |
| Infant, ≤ 14 Days | NA | NA | 20.0 to 25.0 mg/dL | > 25.0 mg/dL |
| (hemolytic) | | | 342 to 428 μmol/L | > 428 μmol/L |
| Blood Urea Nitrogen | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Hyperuricemia | >ULN to 10.0 mg/dL | > 10.0 to 12.0 mg/dL | > 12.0 to 15.0 mg/dL | > 15.0 mg/dL |
| | >ULN to 597 μmol/L | > 597 to 716 μmol/L | > 716 to 895 μmol/L | > 895 μmol/L |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypouricemia | 1.5 mg/dL to < LLN | 1.0 to < 1.5 mg/dL | 0.5 to < 1.0 mg/dL | < 0.5 mg/dL |
| | $87 \mu mol/L$ to $< LLN$ | 57 to < 87 μmol/L | 27 to < 57 μmol/L | < 27 μmol/L |
| Creatinine | > 1.50 to 2.00 mg/dL | > 2.00 to 3.00 mg/dL | > 3.00 to 6.00 mg/dL | > 6.00 mg/dL |
| | > 133 to 177 μmol/L | > 177 to 265 μmol/L | > 265 to 530 μmol/L | > 530 μmol/L |
| Bicarbonate | 16.0 mEq/L to < LLN | 11.0 to < 16.0 mEq/L | 8.0 to < 11.0 mEq/L | < 8.0 mEq/L |
| | 16.0 mmol/L to < LLN | 11.0 to < 16.0 mmol/L | 8.0 to < 11.0 mmol/L | < 8.0 mmol/L |
| Triglycerides | NA | 500 to 750 mg/dL | > 750 to 1200 mg/dL | > 1200 mg/dL |
| (Fasting) | | 5.64–8.47 mmol/L | > 8.47–13.55 mmol/L | > 13.55 mmol/L |
| LDL | 130 to 160 mg/dL | >160 to 190 mg/dL | > 190 mg/dL | NA |
| (Fasting) | 3.35 to 4.15 mmol/L | >4.15 to 4.92 mmol/L | >4.92 mmol/L | |
| Pediatric >2 to <18 years | 110 to 130 mg/dL | >130 to 190 mg/dL | > 190 mg/dL | NA |
| | 2.84 to 3.37 mmol/L | >3.37 to 4.92 mmol/L | >4.92 mmol/L | |
| Hypercholesterolemia | 200 to 239 mg/dL | > 239 to 300 mg/dL | > 300 mg/dL | NA |
| (Fasting) | 5.16 to 6.19 mmol/L | > 6.19 to 7.77 mmol/L | > 7.77 mmol/L | |
| Pediatric < 18 Years | 170 to 199 mg/dL | > 199 to 300 mg/dL | > 300 mg/dL | NA |
| | 4.39 to 5.15 mmol/L | > 5.15 to 7.77 mmol/L | > 7.77 mmol/L | |
| Creatine Kinase | $3.0 \text{ to} < 6.0 \times \text{ULN}$ | 6.0 to < 10.0 × ULN | 10.0 to < 20.0 × ULN | ≥ 20.0 × ULN |

<sup>\*</sup> Calcium should be corrected for albumin if albumin is < 4.0 g/dL

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| ALT (SGPT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| GGT | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Alkaline Phosphatase | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Total Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Pancreatic Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Lipase | > 1.0 to 1.5 × ULN | > 1.5 to 3.0 × ULN | > 3.0 to 5.0 × ULN | > 5.0 × ULN |
| Albumin | 3.0 g/dL to < LLN | 2.0 to < 3.0 g/dL | < 2.0 g/dL | NA |
| | 30 g/L to < LLN | 20 to < 30 g/L | < 20 g/L | |

| URINALYSIS | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hematuria (Dipstick) | 1+ | 2+ | 3-4+ | NA |
| Hematuria (Quantitative) | | | | |
| See Note below | | | | |
| Females | >ULN - 10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Males | 6-10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Proteinuria (Dipstick) | 1+ | 2–3+ | 4+ | NA |
| Proteinuria, 24 Hour Collection | | | | |
| Adult and Pediatric<br>≥ 10 Years | 200 to 999 mg/24 h | >999 to 1999 mg/24 h | >1999 to 3500 mg/24 h | > 3500 mg/24 h |
| Pediatric > 3 Mo to<br>< 10 Years | 201 to 499 mg/m <sup>2</sup> /24 h | >499 to 799 mg/m <sup>2</sup> /24 h | >799 to 1000 mg/m <sup>2</sup> /24 h | > 1000 mg/ m <sup>2</sup> /24 h |
| Glycosuria (Dipstick) | 1+ | 2-3+ | 4+ | NA |

#### Notes:

Toxicity grades for Quantitative and Dipstick Hematuria will be assigned by Covance Laboratory, however for other laboratories, toxicity grades will only be assigned to Dipstick Hematuria.

With the exception of lipid tests, any graded laboratory test with a result that is between the LLN and ULN should be assigned Grade 0.

If the severity of a clinical AE could fall under either one of two grades (e.g., the severity of an AE could be either Grade 2 or Grade 3), select the higher of the two grades for the AE.

| | CARDIOVASCULAR | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cardiac Arrhythmia (general) (By ECG or physical exam) | Asymptomatic AND No intervention indicated | Asymptomatic AND Non-<br>urgent medical intervention<br>indicated | Symptomatic, non-life-<br>threatening AND Non-<br>urgent medical intervention<br>indicated | Life-threatening arrhythmia OR Urgent intervention indicated |
| Cardiac-ischemia/Infarction | NA | NA | Symptomatic ischemia (stable angina) OR Testing consistent with ischemia | Unstable angina OR Acute myocardial infarction |
| Hemorrhage (significant acute blood loss) | NA | Symptomatic AND No transfusion indicated | Symptomatic AND Transfusion of ≤ 2 units packed RBCs (for children ≤ 10 cc/kg) indicated | Life-threatening hypotension<br>OR Transfusion of > 2 units<br>packed RBCs indicated (for<br>children ≤ 10 cc/kg) indicated |
| Hypertension (with repeat testing at same visit) | 140–159 mmHg systolic<br>OR<br>90–99 mmHg diastolic | > 159–179 mmHg systolic<br>OR<br>> 99–109 mmHg diastolic | > 179 mmHg systolic<br>OR<br>> 109 mmHg diastolic | Life-threatening consequences (eg, malignant hypertension) OR Hospitalization (other than ER visit) indicated |
| Pediatric ≤ 17 Years (with repeat testing at same visit) | NA | 91st–94th percentile adjusted<br>for age, height, and gender<br>(systolic and/or diastolic) | ≥ 95th percentile adjusted<br>for age, height, and gender<br>(systolic and/or diastolic) | Life-threatening consequences<br>(eg, malignant hypertension)<br>OR Hospitalization indicated<br>(other than emergency room<br>visit) |
| Hypotension | NA | Symptomatic, corrected with oral fluid replacement | Symptomatic, IV fluids indicated | Shock requiring use of vasopressors or mechanical assistance to maintain blood pressure |
| Pericardial Effusion | Asymptomatic, small effusion requiring no intervention | Asymptomatic, moderate or larger effusion requiring no intervention | Effusion with non-life-<br>threatening physiologic<br>consequences OR Effusion<br>with nonurgent intervention<br>indicated | Life-threatening consequences<br>(eg, tamponade) OR Urgent<br>intervention indicated |

| | | CARDIOVASCULAR | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Prolonged PR Interval | PR interval 0.21 to 0.25 sec | PR interval > 0.25 sec | Type II 2nd degree AV<br>block OR Ventricular pause<br>> 3.0 sec | Complete AV block |
| Pediatric ≤ 16 Years | 1st degree AV block<br>(PR > normal for age and rate) | Type I 2nd degree AV block | Type II 2nd degree AV block | Complete AV block |
| Prolonged QTc | Asymptomatic, QTc interval 0.45 to 0.47 sec OR Increase interval < 0.03 sec above baseline | Asymptomatic, QTc interval 0.48 to 0.49 sec OR Increase in interval 0.03 to 0.05 sec above baseline | Asymptomatic, QTc interval ≥ 0.50 sec OR Increase in interval ≥ 0.06 sec above baseline | Life-threatening<br>consequences, eg, Torsade de<br>pointes or other associated<br>serious ventricular<br>dysrhythmia |
| Pediatric ≤ 16 Years | Asymptomatic, QTc interval 0.450 to 0.464 sec | Asymptomatic, QTc interval 0.465 to 0.479 sec | Asymptomatic, QTc interval ≥ 0.480 sec | Life-threatening consequences, eg, Torsade de pointes or other associated serious ventricular dysrhythmia |
| Thrombosis/Embolism | NA | Deep vein thrombosis AND<br>No intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Deep vein thrombosis AND<br>Intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Embolic event (eg, pulmonary embolism, life-threatening thrombus) |
| Vasovagal Episode (associated with a procedure of any kind) | Present without loss of consciousness | Present with transient loss of consciousness | NA | NA |
| Ventricular Dysfunction<br>(congestive heart failure,<br>CHF) | NA | Asymptomatic diagnostic finding AND intervention indicated | New onset with symptoms<br>OR Worsening symptomatic<br>CHF | Life-threatening CHF |

| RESPIRATORY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Bronchospasm (acute) | FEV1 or peak flow reduced to 70% to 80% | FEV1 or peak flow 50% to 69% | FEV1 or peak flow 25% to 49% | Cyanosis OR FEV1 or peak flow < 25% OR Intubation |
| Dyspnea or Respiratory<br>Distress | Dyspnea on exertion with no or minimal interference with usual social & functional activities | Dyspnea on exertion causing greater than minimal interference with usual social & functional activities | Dyspnea at rest causing inability to perform usual social & functional activities | Respiratory failure with ventilatory support indicated |
| Pediatric < 14 Years | Wheezing OR minimal increase in respiratory rate for age | Nasal flaring OR Intercostal retractions OR Pulse oximetry 90% to 95% | Dyspnea at rest causing inability to perform usual social & functional activities OR Pulse oximetry < 90% | Respiratory failure with ventilatory support indicated |

| | OCULAR/VISUAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Uveitis | Asymptomatic but detectable on exam | Symptomatic anterior uveitis OR Medical intervention indicated | Posterior or pan-uveitis OR<br>Operative intervention<br>indicated | Disabling visual loss in affected eye(s) |
| Visual Changes (from baseline) | Visual changes causing no or minimal interference with usual social & functional activities | Visual changes causing greater than minimal interference with usual social & functional activities | Visual changes causing inability to perform usual social & functional activities | Disabling visual loss in affected eye(s) |

| | | SKIN | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alopecia | Thinning detectable by study participant or caregiver (for disabled adults) | Thinning or patchy hair loss detectable by health care provider | Complete hair loss | NA |
| Cutaneous Reaction – Rash | Localized macular rash | Diffuse macular,<br>maculopapular, or<br>morbilliform rash OR Target<br>lesions | Diffuse macular,<br>maculopapular, or morbilliform<br>rash with vesicles or limited<br>number of bullae OR<br>Superficial ulcerations of<br>mucous membrane limited to<br>one site | Extensive or generalized<br>bullous lesions OR<br>Stevens-Johnson syndrome<br>OR Ulceration of mucous<br>membrane involving two<br>or more distinct mucosal<br>sites OR Toxic epidermal<br>necrolysis (TEN) |
| Hyperpigmentation | Slight or localized | Marked or generalized | NA | NA |
| Hypopigmentation | Slight or localized | Marked or generalized | NA | NA |
| Pruritis (itching – no skin lesions) (See also Injection Site Reactions: Pruritis associated with injection) | Itching causing no or<br>minimal interference with<br>usual social & functional<br>activities | Itching causing greater than minimal interference with usual social & functional activities | Itching causing inability to perform usual social & functional activities | NA |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Anorexia | Loss of appetite without decreased oral intake | Loss of appetite associated with decreased oral intake without significant weight loss | Loss of appetite associated with significant weight loss | Life-threatening consequences<br>OR Aggressive intervention<br>indicated [eg, tube feeding or<br>total parenteral nutrition] |
| Ascites | Asymptomatic | Symptomatic AND Intervention indicated (eg, diuretics or therapeutic paracentesis) | Symptomatic despite intervention | Life-threatening consequences |
| Cholecystitis | NA | Symptomatic AND Medical intervention indicated | Radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences (eg, sepsis or perforation) |
| Constipation | NA | Persistent constipation requiring regular use of dietary modifications, laxatives, or enemas | Obstipation with manual evacuation indicated | Life-threatening consequences (eg, obstruction) |
| Diarrhea | | | | |
| Adult and Pediatric<br>≥1 Year | Transient or intermittent episodes of unformed stools OR Increase of ≤ 3 stools over baseline/24 hr | Persistent episodes of unformed to watery stools OR Increase of 4–6 stools over baseline per 24 hrs. | Bloody diarrhea OR Increase<br>of ≥ 7 stools per 24-hour<br>period OR IV fluid<br>replacement indicated | Life-threatening consequences (eg, hypotensive shock) |
| Pediatric < 1 Year | Liquid stools (more unformed than usual) but usual number of stools | Liquid stools with increased<br>number of stools OR Mild<br>dehydration | Liquid stools with moderate dehydration | Liquid stools resulting in<br>severe dehydration with<br>aggressive rehydration<br>indicated OR Hypotensive<br>shock |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Dysphagia-Odynophagia | Symptomatic but able to eat usual diet | Symptoms causing altered dietary intake without medical intervention indicated | Symptoms causing severely altered dietary intake with medical intervention indicated | Life-threatening reduction in oral intake |
| Mucositis/Stomatitis<br>(clinical exam) See also Proctitis,<br>Dysphagia-Odynophagia | Erythema of the mucosa | Patchy pseudomembranes or ulcerations | Confluent pseudomembranes or ulcerations OR Mucosal bleeding with minor trauma | Tissue necrosis OR Diffuse<br>spontaneous mucosal bleeding<br>OR Life-threatening<br>consequences (eg, aspiration,<br>choking) |
| Nausea | Transient (< 24 hours) or intermittent nausea with no or minimal interference with oral intake | Persistent nausea resulting in decreased oral intake for 24–48 hours | Persistent nausea resulting in minimal oral intake for > 48 hours OR Aggressive rehydration indicated (eg, IV fluids) | Life-threatening consequences (eg, hypotensive shock) |
| Pancreatitis | NA | Symptomatic AND<br>Hospitalization not indicated<br>(other than ER visit) | Symptomatic AND<br>Hospitalization indicated<br>(other than ER visit) | Life-threatening consequences (eg, sepsis, circulatory failure, hemorrhage) |
| Proctitis (functional-<br>symptomatic) Also see Mucositis/<br>Stomatitis for Clinical<br>Exam | Rectal discomfort AND No intervention indicated | Symptoms causing greater than minimal interference with usual social & functional activities OR Medical intervention indicated | Symptoms causing inability to perform usual social/ functional activities OR Operative intervention indicated | Life-threatening consequences (eg, perforation) |
| Vomiting | Transient or intermittent vomiting with no or minimal interference with oral intake | Frequent episodes of vomiting with no or mild dehydration | Persistent vomiting resulting in orthostatic hypotension OR Aggressive rehydration indicated | Life-threatening consequences (eg, hypotensive shock) |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alteration in Personality-<br>Behavior or in Mood (eg,<br>agitation, anxiety,<br>depression, mania,<br>psychosis) | Alteration causing no or minimal interference with usual social & functional activities | Alteration causing greater than minimal interference with usual social & functional activities | Alteration causing inability to perform usual social & functional activities | Behavior potentially harmful<br>to self or others (eg,<br>suicidal/homicidal ideation or<br>attempt, acute psychosis) OR<br>Causing inability to perform<br>basic self-care functions |
| Altered Mental Status For Dementia, see Cognitive and Behavioral/Attentional Disturbance (including dementia and ADD) | Changes causing no or minimal interference with usual social & functional activities | Mild lethargy or somnolence causing greater than minimal interference with usual social & functional activities | Confusion, memory impairment, lethargy, or somnolence causing inability to perform usual social & functional activities | Delirium OR obtundation, OR coma |
| Ataxia | Asymptomatic ataxia detectable on exam OR Minimal ataxia causing no or minimal interference with usual social & functional activities | Symptomatic ataxia causing greater than minimal interference with usual social & functional activities | Symptomatic ataxia causing inability to perform usual social & functional activities | Disabling ataxia causing inability to perform basic self-care functions |
| Cognitive and Behavioral/Attentional Disturbance (including dementia and Attention Deficit Disorder) | Disability causing no or<br>minimal interference with<br>usual social & functional<br>activities OR Specialized<br>resources not indicated | Disability causing greater than minimal interference with usual social & functional activities OR Specialized resources on part-time basis indicated | Disability causing inability to perform usual social & functional activities OR Specialized resources on a full-time basis indicated | Disability causing inability to perform basic self-care functions OR Institutionalization indicated |
| CNS Ischemia (acute) | NA | NA | Transient ischemic attack | Cerebral vascular accident (CVA, stroke) with neurological deficit |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Developmental delay – Pediatric ≤ 16 Years | Mild developmental delay,<br>either motor or cognitive, as<br>determined by comparison<br>with a developmental<br>screening tool appropriate<br>for the setting | Moderate developmental<br>delay, either motor or<br>cognitive, as determined by<br>comparison with a<br>developmental screening tool<br>appropriate for the setting | Severe developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Developmental regression,<br>either motor or cognitive, as<br>determined by comparison<br>with a developmental<br>screening tool appropriate for<br>the setting |
| Headache | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Hospitalization indicated (other than ER visit) OR Headache with significant impairment of alertness or other neurologic function |
| Insomnia | NA | Difficulty sleeping causing greater than minimal interference with usual social/functional activities | Difficulty sleeping causing inability to perform usual social & functional activities | Disabling insomnia causing inability to perform basic self-care functions |
| Neuromuscular Weakness<br>(including myopathy &<br>neuropathy) | Asymptomatic with decreased strength on exam OR Minimal muscle weakness causing no or minimal interference with usual social & functional activities | Muscle weakness causing greater than minimal interference with usual social & functional activities | Muscle weakness causing inability to perform usual social & functional activities | Disabling muscle weakness causing inability to perform basic self-care functions OR Respiratory muscle weakness impairing ventilation |
| Neurosensory Alteration<br>(including paresthesia and<br>painful neuropathy) | Asymptomatic with sensory alteration on exam or minimal paresthesia causing no or minimal interference with usual social & functional activities | Sensory alteration or<br>paresthesia causing greater<br>than minimal interference with<br>usual social & functional<br>activities | Sensory alteration or<br>paresthesia causing inability to<br>perform usual social &<br>functional activities | Disabling sensory alteration or<br>paresthesia causing inability to<br>perform basic self-care<br>functions |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Seizure: (new onset) | NA | 1 seizure | 2–4 seizures | Seizures of any kind that are prolonged, repetitive (eg, status epilepticus), or difficult to control (eg, refractory epilepsy) |
| Seizure: (pre-existing) For Worsening of Existing Epilepsy the Grades Should Be Based on an Increase from Previous Level of Control to Any of These Levels | NA | Increased frequency of pre-<br>existing seizures (non-<br>repetitive) without change in<br>seizure character OR<br>infrequent breakthrough<br>seizures while on stable meds<br>in a previously controlled<br>seizure disorder | Change in seizure character<br>from baseline either in<br>duration or quality (eg,<br>severity or focality) | Seizures of any kind that are prolonged, repetitive (eg, status epilepticus), or difficult to control (eg, refractory epilepsy) |
| Seizure - Pediatric < 18 Years | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>< 5 minutes with < 24 hours<br>post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting 5–20<br>minutes with<br>< 24 hours post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>> 20 minutes | Seizure, generalized onset<br>with or without secondary<br>generalization, requiring<br>intubation and sedation |
| Syncope (not associated with a procedure) | NA | Present | NA | NA |
| Vertigo | Vertigo causing no or<br>minimal interference with<br>usual social & functional<br>activities | Vertigo causing greater than minimal interference with usual social & functional activities | Vertigo causing inability to perform usual social & functional activities | Disabling vertigo causing inability to perform basic self-care functions |

| | MUSCULOSKELETAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Arthralgia See also Arthritis | Joint pain causing no or minimal interference with usual social & functional activities | Joint pain causing greater than minimal interference with usual social & functional activities | Joint pain causing inability to perform usual social & functional activities | Disabling joint pain causing inability to perform basic self-care functions |
| Arthritis See also Arthralgia | Stiffness or joint swelling causing no or minimal interference with usual social & functional activities | Stiffness or joint swelling causing greater than minimal interference with usual social & functional activities | Stiffness or joint swelling causing inability to perform usual social & functional activities | Disabling joint stiffness or<br>swelling causing inability to<br>perform basic self-care<br>functions |
| Bone Mineral Loss | BMD t-score or z-score<br>-2.5 to -1.0 | BMD t-score or z-score < -2.5 | Pathological fracture<br>(including loss of vertebral<br>height) | Pathologic fracture causing life-threatening consequences |
| Pediatric < 21 Years | BMD z-score<br>-2.5 to -1.0 | BMD z-score < -2.5 | Pathological fracture<br>(including loss of vertebral<br>height) | Pathologic fracture causing life-threatening consequences |
| Myalgia<br>(non-injection site) | Muscle pain causing no or minimal interference with usual social & functional activities | Muscle pain causing greater than minimal interference with usual social & functional activities | Muscle pain causing inability to perform usual social & functional activities | Disabling muscle pain causing inability to perform basic self-care functions |
| Osteonecrosis | NA | Asymptomatic with radiographic findings AND No operative intervention indicated | Symptomatic bone pain with radiographic findings OR Operative intervention indicated | Disabling bone pain with radiographic findings causing inability to perform basic self-care functions |

| | SYSTEMIC | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Acute Systemic Allergic<br>Reaction | Localized urticaria<br>(wheals) with no medical<br>intervention indicated | Localized urticaria with medical intervention indicated OR Mild angioedema with no medical intervention indicated | Generalized urticaria OR<br>Angioedema with medical<br>intervention indicated OR<br>Symptomatic mild<br>bronchospasm | Acute anaphylaxis OR Life-<br>threatening bronchospasm OR<br>laryngeal edema |
| Chills | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Fatigue<br>Malaise | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Incapacitating fatigue/malaise symptoms causing inability to perform basic self-care functions |
| Fever (nonaxillary) | 37.7°C to 38.6°C<br>99.8°F to 101.5°F | 38.7°C to 39.3°C<br>101.6°F to 102.8°F | 39.4°C to 40.5°C<br>102.9°F to 104.9°F | > 40.5°C<br>> 104.9°F |
| Pain- Indicate Body Site See also Injection Site Pain, Headache, Arthralgia, and Myalgia | Pain causing no or<br>minimal interference with<br>usual social & functional<br>activities | Pain causing greater than minimal interference with usual social & functional activities | Pain causing inability to perform usual social & functional activities | Disabling pain causing inability to perform basic self-care functions OR Hospitalization (other than ER visit) indicated |
| Unintentional Weight<br>Loss | NA | 5% to 9% loss in body weight from baseline | 10% to 19% loss in body weight from baseline | ≥ 20% loss in body weight<br>from baseline OR Aggressive<br>intervention indicated [eg,<br>tube feeding or total parenteral<br>nutrition] |

| | INJECTION SITE REACTION | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Injection Site Pain (pain without touching) Or Tenderness (pain when area is touched) | Pain/tenderness causing no or minimal limitation of use of limb | Pain/tenderness limiting use of limb OR Pain/tenderness causing greater than minimal interference with usual social & functional activities | Pain/tenderness causing inability to perform usual social & functional activities | Pain/tenderness causing inability<br>to perform basic self-care<br>function OR Hospitalization<br>(other than ER visit) indicated<br>for management of<br>pain/tenderness |
| Injection Site Reaction (Localized), > 15 Years | Erythema OR Induration<br>of $5 \times 5$ cm to $9 \times 9$ cm (or<br>$25-81 \times \text{cm}^2$ ) | Erythema OR Induration OR<br>Edema > 9 cm any diameter<br>(or > 81 cm <sup>2</sup> ) | Ulceration OR Secondary<br>infection OR Phlebitis OR<br>Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pediatric ≤ 15 Years | Erythema OR Induration<br>OR Edema present but<br>≤ 2.5 cm diameter | Erythema OR Induration<br>OR Edema > 2.5 cm<br>diameter but < 50% surface<br>area of the extremity<br>segment (eg, upper<br>arm/thigh) | Erythema OR Induration OR Edema involving ≥ 50% surface area of the extremity segment (eg, upper arm/thigh) OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pruritis Associated with Injection See also Skin: Pruritis (itching—no skin lesions) | Itching localized to injection<br>site AND Relieved<br>spontaneously or with<br>< 48 h treatment | Itching beyond the injection site but not generalized OR Itching localized to injection site requiring ≥ 48 h treatment | Generalized itching causing inability to perform usual social & functional activities | NA |

| | ENDOCRINE/METABOLIC | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Lipodystrophy (eg, back of neck, breasts, abdomen) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious changes on casual visual inspection | NA |
| Diabetes Mellitus | NA | New onset without need to initiate<br>medication OR Modification of<br>current meds to regain glucose<br>control | New onset with initiation of indicated med OR Diabetes uncontrolled despite treatment modification | Life-threatening consequences<br>(eg, ketoacidosis,<br>hyperosmolar non-ketotic<br>coma) |
| Gynecomastia | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |
| Hyperthyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid suppression therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, thyroid storm) |
| Hypothyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid replacement therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, myxedema coma) |
| Lipoatrophy (eg, fat loss from the face, extremities, buttocks) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |

| | | GENITOURINARY | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Intermenstrual Bleeding (IMB) | Spotting observed by participant OR Minimal blood observed during clinical or colposcopic exam | Intermenstrual bleeding not greater in duration or amount than usual menstrual cycle | Intermenstrual bleeding greater in duration or amount than usual menstrual cycle | Hemorrhage with life-<br>threatening hypotension OR<br>Operative intervention<br>indicated |
| Urinary Tract obstruction (eg, stone) | NA | Signs or symptoms of urinary tract obstruction without hydronephrosis or renal dysfunction | Signs or symptoms of urinary tract obstruction with hydronephrosis or renal dysfunction | Obstruction causing life-<br>threatening consequences |

| | | INFECTION | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Infection (any other than HIV infection) | Localized, no systemic antiµbial treatment indicated AND Symptoms causing no or minimal interference with usual social & functional activities | Systemic antiµbial treatment indicated OR Symptoms causing greater than minimal interference with usual social & functional activities | Systemic antiubial treatment indicated AND Symptoms causing inability to perform usual social & functional activities OR Operative intervention (other than simple incision and drainage) indicated | Life-threatening consequences (eg, septic shock) |

Basic Self-care Functions: Activities such as bathing, dressing, toileting, transfer/movement, continence, and feeding.

Usual Social & Functional Activities: Adaptive tasks and desirable activities, such as going to work, shopping, cooking, use of transportation, pursuing a hobby, etc

# Appendix 4. Tanner Stages

| | 1. Pubic hair (male and female) |
|---|---|
| Tanner I | no pubic hair at all (prepubertal Dominic state) |
| Tanner II | small amount of long, downy hair with slight pigmentation at the base of the penis and scrotum (males) or on the labia majora (females) |
| Tanner III | hair becomes more coarse and curly, and begins to extend laterally |
| Tanner IV | adult-like hair quality, extending across pubis but sparing medial thighs |
| Tanner V | hair extends to medial surface of the thighs |
| | 2. Genitals (male) (One standard deviation around mean age) |
| Tanner I | Testes, scrotum, and penis about same size and proportion as in early childhood |
| Tanner II | Enlargement of scrotum and testes; skin of scrotum reddens and changes in texture; little or no enlargement of penis (10.5-12.5) |
| Tanner III | Enlargement of penis, first mainly in length; further growth of testes and scrotum (11.5-14) |
| Tanner IV | Increased size of penis with growth in breadth and development of glans; further enlargement of testes and scrotum and increased darkening of scrotal skin (13.5-15) |
| Tanner V | Genitalia adult in size and shape |
| | 3. Breasts (female) |
| Tanner I | no glandular tissue: areola follows the skin contours of the chest |
| Tanner II | breast bud forms, with small area of surrounding glandular tissue; areola begins to widen |
| Tanner III | breast begins to become more elevated, and extends beyond the borders of the areola, which continues to widen but remains in contour with surrounding breast |
| Tanner IV | increased breast size and elevation; areola and papilla form a secondary mound projecting from the contour of the surrounding breast |
| Tanner V | breast reaches final adult size; areola returns to contour of the surrounding breast, with a projecting central papilla. |

# Appendix 5. Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements

### 1. Background

RBV is contraindicated in pregnancy as significant teratogenic and embryocidal effects have been demonstrated in all animal species tested. Pregnancy must be excluded before the start of treatment with study drugs and prevented thereafter by reliable contraceptive methods. Pregnancy tests will be performed regularly throughout this study. Furthermore, RBV is known to accumulate intracellularly where it is cleared slowly, and is also excreted in semen. Therefore, extreme care must be taken to avoid pregnancy during RBV therapy and for up to 6 months following completion of treatment (7 months for males). Please refer to the latest version of the product insert for additional information.

Non-clinical toxicity studies of sofosbuvir demonstrated no adverse effect on fertility or embryo-fetal development. However, there are no clinical studies of sofosbuvir in pregnant women. Please refer to the latest version of the investigator's brochure for additional information.

# 2. Definition of Female of Childbearing Potential and Contraceptive Requirements for Female Subjects (and their male partners)

For the purpose of this trial, all post-menarchal females will be considered to be of childbearing potential, unless there is documentation of irreversible ovarian failure or surgical sterilization.

Post menarchal females must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on the Day 1 visit prior to randomization. They must also agree to one of the following from 3 weeks prior to Day 1 until 6 months after last dose of RBV:

• Complete abstinence from intercourse. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

Or

- Consistent and correct use of 1 of the following methods of birth control listed below, in addition to a male partner who correctly uses a condom, from the date of Screening until 6 months after the last dose of RBV:
  - intrauterine device (IUD) with a failure rate of < 1% per year
  - female barrier method: cervical cap or diaphragm with spermicidal agent
  - tubal sterilization
  - vasectomy in male partner

- implants of levonorgestrel
- injectable progesterone
- oral contraceptives (either combined or progesterone only)
- contraceptive vaginal ring
- transdermal contraceptive patch

# 3. Contraceptive Requirements for Male Subjects (and their female partners)

All male study participants must agree to consistently and correctly use a condom from Baseline until 7 months after the last dose of RBV. If their female partner is of childbearing potential (as defined above), their female partner must use 1 of the methods of birth control listed above from the date of Screening until 7 months after last dose of RBV.

Male subjects must agree to refrain from sperm donation for at least 7 months after the last dose of RBV.

## 4. Procedures to be Followed in the Event of Pregnancy

Subjects will be instructed to notify the investigator if they become pregnant at any time during the study, or if they become pregnant within 6 months (7 months for partners of male subjects) of last RBV dose. Subjects who become pregnant or who suspect that they are pregnant must report the information to the investigator and discontinue study drug immediately. Subjects whose partner has become pregnant or suspects she is pregnant must report the information to the investigator.

Instructions for reporting pregnancy, partner pregnancy, and pregnancy outcome are outlined in Section 8.5.2.1.